



# **CLINICAL PROTOCOL**

# A 12-Week, Randomised, Controlled, Examiner-blind, Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste for the Relief of Dentine Hypersensitivity in a Chinese Population

| Protocol Number: | 300026 |
|---|---|
| Compound/Product Name: | Stannous fluoride (SnF <sub>2</sub> ) |
| United States (US) Investigational<br>New Drug (IND) Number: | Not Applicable (N/A) |
| European Clinical Trials Database (EudraCT) Number: | N/A |
| Other Regulatory Agency Identified Number: | N/A |
| Phase: | N/A |

This document contains confidentiality statements that are not relevant for this publicly available version

Protocol Number: 300026



# **Sponsor Information**

| Sponsor Name & Legal<br>Registered Address | GlaxoSmithKline Consumer Healthcare (UK) Trading Limited |
|---|---|
| | St Georges Avenue, |
| | Weybridge, |
| | Surrey, |
| | KT13 0DE, |
| | United Kingdom (UK) |
| Sponsor Contact Details | GlaxoSmithKline Consumer Healthcare (GSK CH) |
| | 25/F and 26/F, No.90 QirongRoad, Pudong New Area, Shanghai, China |
| | Tel: 021-2301 9366 |

Protocol Number: 300026



# **Document History**

| Document | Version | Summary of Changes |
|---|---|---|
| Original protocol | 1.0 | N/A |
| Amendment 1 | 2.0 | Minor amendment: In section 6.5, clarification on the blinding has been added as following: "As a matter of study conduct, including emergency unblinding events, only the investigator may learn the contents of one or more of the product codes used to allocate study product, not the clinical examiners. Given the application of IRT within this study, any such knowledge will not affect the decision to enroll a subject or influence the order in which subjects are enrolled" |
| Amendment 2 | 3.0 | Minor amendments: 1) Sponsor address in China has been updated 2) Section 5.1 Type and planned number of subjects, the sentence "their use would not be expected to cause harm to the mother, the foetus or baby" has been deleted for clarification 3) In section 10, the safety email inbox has been amended from PPD to PPD |

Amendments incorporate all revisions to date, including amendments made at the request of country health authorities, institutional review boards/ethics committees (IRBs/ECs), etc.





# **Principal Investigator Protocol Agreement Page**

- I confirm agreement to conduct the study in compliance with the protocol and any amendments according to the current International Conference on Harmonisation Good Clinical Practice (ICH GCP) guidelines.
- I acknowledge that I am responsible for overall study conduct. I agree to personally conduct or supervise the described study.
- I agree to ensure that all associates, colleagues and employees assisting in the conduct of the study are informed about their obligations. Mechanisms are in place to ensure site staff receives all appropriate information throughout the study.
- I agree to conduct this study in full conformance with the laws and regulations of the country in which the research is conducted and the Declaration of Helsinki.

| Investigator Name: | PPD |
|------------------------------|-----|
| Investigator Qualifications: | PPD |
| Investigator Signature: | PPD |
| Date of Signature/Agreement: | PPD |

Clinical Protocol

Protocol Number: 300026



| Та | | f Conte | | _ |
|----|-----------|-----------|----------------------------------|----|
| | _ | | nation | |
| | | | tory | |
| | | _ | stigator Protocol Agreement Page | |
| | | | ents | |
| 1 | | | SUMMARY | |
| | 1.1 | • • | iis | |
| | 1.2 | | lle of Activities | |
| 2 | | | ION | |
| | 2.1 | • | Rationale and Background | |
| | 2.2 | | t/Risk Assessment | |
| | 2.3 | | nism of Action/Indication | |
| 3 | | | ECTIVES AND ENDPOINTS | |
| 4 | STUI | DY DESI | GN | 17 |
| | 4.1 | Overall | l Design | 17 |
| | 4.2 | Scientif | fic Rationale for Study Design | 18 |
| | 4.3 | Justifica | ation for Dose | 20 |
| | 4.4 | End of | Study Definition | 21 |
| 5 | STUI | OY POPU | JLATION | 21 |
| | 5.1 | Type ar | nd Planned Number of Subjects | 21 |
| | 5.2 | Inclusio | on Criteria | 22 |
| | 5.3 | Exclusi | ion Criteria | 23 |
| | 5.4 | Randon | mization Criteria | 25 |
| | 5.5 | Lifestyl | le Considerations | 25 |
| | | 5.5.1 | Oral Care Restrictions | 26 |
| | | 5.5.2 | Dietary and Alcohol Restrictions | 26 |
| | | 5.5.3 | Covid-19 | |
| | | 5.5.4 | Contraception | 26 |
| | 5.6 | Screen | Failures | |
| | 5.7 | Sponso | or's Qualified Medical Personnel | 27 |
| | 5.8 | _ | al Assessor Qualifications | |
| 6 | STUI | | DUCTS | |
| | 6.1 | | Product Supplies | |
| | | 6.1.1 | Dosage Form and Packaging | |
| | | 6.1.2 | Product Dispensing | |
| | 6.2 | | istration | |
| | ~ <b></b> | 6.2.1 | Product Dosing Errors | |
| | | 6.2.2 | Overdose | |
| | 6.3 | | Product Storage | |
| | 0.0 | ~~~, 1 | | |

# Clinical Protocol

# Protocol Number: 300026



| | 6.4 | Study Pr | oduct Accountability | 32 |
|---|---|---|---|---|
| | | 6.4.1 | Destruction of Study Product Supplies | |
| | 6.5 | Blinding | and Allocation/Randomization | |
| | 6.6 | Breaking | g the Blind | 33 |
| | 6.7 | Complia | nce | 34 |
| | 6.8 | Concom | itant Medications/Treatments | 34 |
| 7 | DISC | CONTINUA | ATION OF STUDY INTERVENTION AND SUBJECT | |
| | DISC | | ATION/WITHDRAWAL | |
| | 7.1 | Subject I | Discontinuation/Withdrawal | 35 |
| | 7.2 | Lost to F | Follow up | 36 |
| 8 | STU | DY PROCI | EDURES | 36 |
| | 8.1 | Visit 1/S | creening | 36 |
| | | 8.1.1 | Informed Consent | 36 |
| | | 8.1.2 | Demographics | 37 |
| | | 8.1.3 | Check of the WeChat Application | 37 |
| | | 8.1.4 | DH Screening Questionnaire | 37 |
| | | 8.1.5 | Review of Oral Care Products | 37 |
| | | 8.1.6 | Review of Brushing Habits | 38 |
| | | 8.1.7 | Medical History and Prior Medication/Treatment | 38 |
| | | 8.1.8 | Clinical Examinations and Assessments | 38 |
| | | 8.1.9 | Inclusion/Exclusion Criteria | 38 |
| | | 8.1.10 | Subject Eligibility | 39 |
| | | 8.1.11 | Supervised Brushing with Acclimatization Toothpaste | 39 |
| | 8.2 | Study Pe | eriod | 39 |
| | | 8.2.1 | Visit 2 (Baseline/Day 1) | 39 |
| | | 8.2.2 | Visit 3 (Week 6/Day 43 $\pm$ 4) and Visit 4 (Week 12/Day 85 $\pm$ 4) | 42 |
| | 8.3 | Study Co | onclusion | 43 |
| | 8.4 | Follow-u | ıp Visit / Phone Call | 43 |
| 9 | STU | DY ASSES | SSMENTS | 43 |
| | 9.1 | Screenin | g Assessments | 44 |
| | | 9.1.2 | Qualifying Tactile Sensitivity | 45 |
| | | 9.1.3 | Qualifying Evaporative (Air) Sensitivity | 46 |
| | 9.2 | Dentine | Hypersensitivity Efficacy Assessments | 47 |
| | | 9.2.1 | Tactile Sensitivity Assessment (Yeaple Probe) | 47 |
| | | 9.2.2 | Evaporative (Air) Sensitivity Assessments | |
| | 9.3 | Safety ar | nd Other Assessments | |
| | | 9.3.1 | Oral Soft Tissue (OST) Examination | |
| | | 9.3.2 | Oral Hard Tissue (OHT) Examination | |
| | | 9.3.3 | Pregnancy | |
| | | | = · · · · · | |



| 10 | ADV | ERSE EV | ENT AND SERIOUS ADVERSE EVENTS | 49 |
|---|---|---|---|---|
| | 10.1 | Definiti | on of an Adverse Event (AE) | 49 |
| | 10.2 | Definiti | on of a Serious Adverse Event (SAE) | 50 |
| | 10.3 | Time Pe | eriod and Frequency for Collecting AE and SAE Information | 51 |
| | 10.4 | Reporti | ng Procedures | 51 |
| | | 10.4.1 | Reporting of an Adverse Event | 52 |
| | | 10.4.2 | Reporting of a Serious Adverse Event | 52 |
| | 10.5 | Evaluat | ing Adverse Events | 53 |
| | | 10.5.1 | Assessment of Intensity | 53 |
| | | 10.5.2 | Assessment of Causality | 53 |
| | 10.6 | Follow- | up of AEs and SAEs | 54 |
| | 10.7 | • | | |
| | 10.8 | Regulat | ory Reporting Requirements for SAEs | 55 |
| | 10.9 | | ıcy | |
| | | 10.9.1 | Time Period for Collecting Pregnancy Information | 55 |
| | | 10.9.2 | Action to be Taken if Pregnancy Occurs | 55 |
| 11 | DATA | A MANA | GEMENT | |
| | 11.1 | Case Re | eport Form | 56 |
| | 11.2 | Data Ha | andling | 57 |
| | | 11.2.1 | Data Queries | 57 |
| 12 | STATISTICAL CONSIDERATIONS AND DATA ANALYSES | | | |
| | 12.1 Sample Size Determination | | | |
| | 12.2 | Populations for Analysis | | |
| | | 12.2.1 | Definitions of Analysis Populations | 58 |
| | | 12.2.2 | Exclusion of Data from Analysis | 58 |
| | 12.3 Statistical Analyses | | | |
| | | 12.3.1 | Primary Analysis | 59 |
| | | 12.3.2 | Secondary Analyses | 59 |
| | | 12.3.3 | Safety Analyses | 60 |
| | | 12.3.4 | Demographic and Baseline Characteristics | 61 |
| | | 12.3.5 | Study Product Compliance and Use of Other Therapies | 61 |
| | | 12.3.6 | Handling of Dropouts and Missing Data | 61 |
| | | 12.3.7 | Interim Analysis | 62 |
| 13 | STUL | Y GOVE | ERNANCE CONSIDERATIONS | 62 |
| | 13.1 Quality Control | | | |
| | 13.2 | Quality | Assurance | 62 |
| | 13.3 Regulatory and Ethical Considerations | | | |
| | | 13.3.1 | Institutional Review Board | 63 |
| | 13.3.2 Ethical Conduct of the Study | | | 63 |
| | | | • | |

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH

# 300026 Protocol Amendment Project Ox 14 Feb 2023 | TMF-238226 | 3.0

# GSK Consumer Healthcare

# Clinical Protocol

# Protocol Number: 300026



| | | 13.3.3 | Subject Information and Consent | 63 |
|---|---|---|---|---|
| | | 13.3.4 | Subject Recruitment | 64 |
| | | 13.3.5 | Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP | 64 |
| | 13.4 | Posting o | f Information on Publicly Available Clinical Trial Registers | 64 |
| | 13.5 | Provision | of Study Results to Investigators | 64 |
| | 13.6 | Records | Retention | 65 |
| | 13.7 | Condition | ns for Terminating the Study | 65 |
| 14 | REFE | RENCES. | | 66 |
| 15 | APPE | NDICES | | 69 |
| | 15.1 | ABBREV | /IATIONS | 69 |
| | 15.2 | Screening | g questionnaire | 71 |
| | 15.3 | Video Co | ompliance Check-list | 73 |

# 300026 Protocol Amendment Project Ox 14 Feb 2023 | TMF-238226 | 3.0

**GSK** Consumer Healthcare

Clinical Protocol

Protocol Number: 300026



# List of in text tables

| Table 1-1 | Schedule of Activities | 13 |
|------------|---------------------------------------------|----|
| Table 3-1 | Study Objectives and Endpoints | 16 |
| Table 4-1 | Eligibility Checks for Test Tooth Selection | 20 |
| Table 6-1 | Study Product Supplies | 28 |
| Table 6-2 | Acclimatization Product | 29 |
| Table 6-3 | Sundry Items | 29 |
| Table 15-1 | Abbreviations | 69 |

Protocol Number: 300026



# 1 PROTOCOL SUMMARY

# 1.1 Synopsis

### **Short Title:**

Randomized Controlled Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Toothpaste for the Relief of Dentine Hypersensitivity in a Chinese Population.

# **Background and Rationale:**

The sponsor markets 0.454% weight/weight (w/w) stannous fluoride (SnF<sub>2</sub>) toothpastes for the relief of dentine hypersensitivity (DH) globally; clinical efficacy is supported by two 8-week DH studies conducted outside China. Chinese Ministry of Health (MoH) guidelines require two clinical studies to support the efficacy of a functional toothpaste; at least one of these studies (for each claimed benefit) must be conducted on a local Chinese population (Ministry of Health China, 2010). Thus, a clinical study conducted in the Chinese population is required to support long-term DH relief claims for 0.454% w/w stannous fluoride (SnF<sub>2</sub>) toothpastes in China.

# **Objectives and Endpoints:**

| Objectives | Endpoints |
|---|---|
| Primary | |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to an evaporative (air) stimulus (as measured by Schiff sensitivity score), compared to a negative control toothpaste, after 12 weeks twice daily use. | Change from Baseline in Schiff sensitivity score at Week 12. |
| Secondary | |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to a tactile stimulus (as measured by tactile threshold), compared to a negative control toothpaste, after 12 weeks twice daily use. | Change from Baseline in tactile threshold (grams [g]) at Week 12. |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to an evaporative (air) stimulus (as measured by Visual Analogue Scale [VAS]), compared to a negative control toothpaste, after 12 weeks twice daily use. | Change from Baseline in VAS (millimeters [mm]) at Week 12. |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to evaporative (air) and tactile stimuli (as measured by Schiff sensitivity score/VAS and tactile threshold, respectively), compared to a negative control toothpaste, after 6 weeks twice daily use. | Change from Baseline in Schiff sensitivity score, tactile threshold (g) and VAS (mm) at Week 6. |
| To determine the clinical efficacy of a 5.0% w/w calcium sodium phosphosilicate (CSPS) toothpaste (positive control) in reducing DH to evaporative (air) and tactile stimuli (as measured by Schiff sensitivity score/VAS and tactile threshold, respectively), compared to a negative control toothpaste, after 6 and 12 weeks twice daily use. | Change from Baseline in Schiff sensitivity score and tactile threshold (g) and VAS (mm) at Week 6 and Week 12. |

Clinical Protocol

Protocol Number: 300026



| Safety | |
|-------------------------------------------------|----------------------------|
| | Treatment emergent adverse |
| toothpastes when used twice daily for 12 weeks. | events (TEAEs) |

# **Study Design:**

This will be a single centre, 12-week, randomized, controlled, examiner-blind, 3 treatment arm, parallel group design, stratified (by maximum Baseline Schiff sensitivity score of the two selected 'test teeth') clinical study, investigating the clinical efficacy of a 0.454% SnF<sub>2</sub> toothpaste for the relief of DH in a Chinese population.

Randomized subjects will be requested to brush their teeth twice daily (morning and evening) with their assigned study toothpaste for the duration of the 12-week study period. DH will be assessed at Screening, Baseline (Day 1), Week 6 and Week 12 using three clinical measures (an evaporative (air) stimulus with Schiff sensitivity score; a tactile stimulus with tactile threshold [g]; an evaporative (air) stimulus with VAS [mm]). Safety and oral tolerability of the study products will be monitored over the 12-week usage period by review of reported adverse events (AEs).

A 5.0% w/w CSPS toothpaste with clinically proven longer term DH efficacy in the Chinese population will be included in the study as a positive control. The clinical efficacy of both antisensitivity toothpastes (test and positive control) will be compared with that of a regular fluoride toothpaste (negative control), with no known anti-sensitivity properties.

### **Study Products:**

| Product<br>Description | Test Toothpaste | Reference Toothpaste<br>(Positive Control) | Reference Toothpaste<br>(Negative Control) |
|---|---|---|---|
| Product Name | 0.454% w/w SnF <sub>2</sub><br>toothpaste | 5.0% w/w CSPS<br>toothpaste | Regular fluoride toothpaste |
| | (Sensodyne Sensitivity & Gum*) | (Sensodyne Repair & Protect*) | (Crest Cavity Protection<br>Fresh Lime*) |
| Master<br>Formulation Code | CCI | CCI | Not applicable (N/A) |
| Fluoride Content | 1100 parts per million (ppm) fluoride as SnF <sub>2</sub> | 1150 ppm fluoride as sodium fluoride (NaF) | 1150 ppm fluoride as<br>NaF |

<sup>\*</sup> Chinese commercial product

# Type and Planned Number of Subjects:

Male and female subjects aged 18-70 years (inclusive), in good general and oral health, with no clinically relevant abnormalities in medical history, or upon oral examination, that could impact subject safety or well-being, or the outcomes of the study. Female subjects who are pregnant, or intending to become pregnant during the study, or breast-feeding, will not be included.

Eligible subjects will have a minimum of 20 natural teeth, a self-reported history of tooth sensitivity and at least two teeth with clinical examiner-confirmed DH (tactile threshold  $\leq$  20 g; Schiff sensitivity score  $\geq$  2) at both Screening and Baseline and VAS  $\geq$  40 mm at Baseline; in addition, the selected test teeth must demonstrate a consistent response to the evaporative (air) stimulus at the Screening and Baseline visits (i.e., Schiff sensitivity score = 2 at Screening and Baseline, **or** Schiff sensitivity score = 3 at Screening and Baseline; <u>Table 4-1</u>).

Clinical Protocol

Protocol Number: 300026



Sufficient subjects will be screened to randomize approximately 240 subjects to study treatment to ensure approximately 235 subjects complete the study (approximately 94 each for test toothpaste and negative control, and 47 for positive control), allowing for approximately 2% dropouts after randomization, as observed in previous clinical studies conducted in China.

### **Statistical Analysis Summary:**

A modified Intent-To-Treat (mITT) population will be used for the efficacy analyses (all randomized subjects who complete at least one use of study product and have at least one post Baseline clinical efficacy assessment).

Schiff sensitivity score, tactile threshold (g) and VAS (mm) will be derived as the average score or value, respectively, of the 2 test teeth (identified at Baseline). Change from Baseline will be derived for the individual teeth first before calculating the average change of the 2 test teeth.

Significance testing will be conducted at the two-sided 5% significance level.

Change from Baseline in Schiff sensitivity score will be analysed using a Mixed Model with Repeated Measures (MMRM) with study product, visit and study product x visit interaction as fixed effects and Baseline Schiff sensitivity score as a covariate. Subject will be included as a repeated measure with unstructured covariance matrix. Kenward Rogers degrees of freedom approach will be applied.

For the primary endpoint (change from Baseline in Schiff sensitivity score at Week 12), the difference between least square means for the test toothpaste compared to the negative control at Week 12 from the MMRM will be presented along with the two-sided p-value and 95% confidence intervals (CIs) to test the primary hypothesis of the study.

Change from Baseline in tactile threshold (g) will be analysed using the same MMRM as the primary endpoint but with Baseline tactile threshold as a covariate, rather than Baseline Schiff sensitivity score. In addition, the maximum Baseline Schiff sensitivity score across test teeth (2 or 3) will be fitted as a fixed effect. The difference between least square means for the test toothpaste compared to the negative control at Week 12 from the MMRM will be presented, along with the two-sided p-value and 95% CIs.

Change from Baseline in VAS (mm) will be analysed using the same MMRM as for the change from Baseline in tactile threshold (g) but with Baseline VAS (mm) as a covariate, rather than the Baseline tactile threshold (g). The difference between least square means for the test toothpaste vs. negative control at Week 12 will be presented, along with the two-sided p-value and 95% CIs.

For the other secondary endpoints, the differences between least square mean change from Baseline from the respective MMRM (test toothpaste vs. negative control at Week 6, positive vs. negative control at Weeks 6 and 12) will be presented with two-sided p-values and 95% CIs.

The assumption of normality and homogeneity of variance in each MMRM will be investigated. In case of violation of these assumptions, a suitable non-parametric test (adjusted for the randomisation stratification) will be performed to assess the change from Baseline comparisons (test toothpaste vs. negative control and positive control vs. negative control at Week 6 and Week 12) and results will be provided to support the MMRM results; the non-parametric results will be considered to supersede the MMRM results under the observation of strong violations of the above assumptions.

Protocol Number: 300026



# 1.2 Schedule of Activities

The schedule of activities table provides an overview of the subject visits and study procedures. The investigator may schedule visits (unplanned visits) in addition to those listed on the schedule of activities, to conduct evaluations or assessments required to protect the well-being of the subject.

Table 1-1 Schedule of Activities

| | Screening | | Study Visits | | |
|---|---|---|---|---|---|
| Procedure/Assessment | Visit 1 | | Visit 2 Baseline (Day 1) | Visit 3<br>Week 6<br>(Day 43±4) | Visit 4<br>Week 12<br>(Day 85±4) |
| Informed consent <sup>1</sup> | X | | | | |
| Demographics | X | | | | |
| Confirm WeChat application available on subject's mobile phone <sup>2</sup> | X | | | | |
| DH screening questionnaire | X | | | | |
| Confirm absence of anti-sensitivity ingredients & DH claims from subject's own oral care products | X | | | | |
| Review subject's normal oral hygiene routine, specifically their rinsing habits | X | | | | |
| Medical history and prior/current medication/treatment review | X | | | | |
| Changes in health and medications/treatments | | \ccl | X | X | X |
| Compliance checks Check returned study supplies, review diary & evaluate compliance with twice daily use. Check compliance with Lifestyle Guidelines/ Medication requirements. | | Acclimatization Period (14-28 Days) | X | X | X |
| Check brushing videos to confirm compliance with acclimatisation toothpaste usage instructions | | iod (12 | X | | |
| Oral soft tissue (OST) examination | X | 1-28 | X | X | X |
| Oral hard tissue (OHT) examination | X | Day | | | X |
| Eligible teeth assessments (dentition exclusions, Erosion/Abrasion/Recession [EAR], Modified Gingival Index [MGI], clinical mobility) | X | /s) | | | |
| Qualifying tactile sensitivity assessment (tactile threshold (g)) for all eligible teeth <sup>3,4</sup> | X | | X | | |
| Qualifying evaporative (air) sensitivity assessments (Schiff sensitivity score, VAS) for all eligible teeth with a tactile threshold $\leq 20 g^{3,4}$ | X | | X | | |
| $\label{eq:linear_constraints} Identify all eligible teeth which qualify for Baseline sensitivity assessments: \\ - No dentition exclusions \\ - Presence of EAR \\ - MGI = 0 adjacent to the test area only \\ - Clinical mobility = 0 \\ - Tactile threshold \leq 20g \\ - Schiff sensitivity score \geq 2$ | X | | | | |

Clinical Protocol

Protocol Number: 300026



| Select two test teeth <sup>5</sup> | | X | | |
|---|---|---|---|---|
| Inclusion/exclusion criteria | X | X | | |
| Subject eligibility | X | X | | |
| Subject continuance | | | X | X |
| Dispense acclimatisation toothpaste, toothbrush, rinsing cups, timer and diary | X | | | |
| Supervised brushing with acclimatisation toothpaste <sup>6</sup> | X | | | |
| Return to site with acclimatisation toothpaste, toothbrush and completed diary | | X | | |
| Stratification and randomisation | | X | | |
| Dispense study toothpaste, toothbrush, rinsing cups and diary | | X | | |
| Dispense toothbrush only | | | X | |
| Supervised brushing with study toothpaste and reminder of product usage instructions <sup>6,7</sup> | | X | X | |
| Return to site with study toothpaste, toothbrush and completed diary | | | X | X |
| Tactile sensitivity assessment (tactile threshold): Two test teeth only <sup>5</sup> | | | X | X |
| Evaporative (air) sensitivity assessment (Schiff sensitivity score, VAS): Two test teeth only <sup>5</sup> | | | X | X |
| Study conclusion | | | | X |
| Monitor adverse events (AEs) <sup>8</sup> | X | X | X | X |

### **Footnotes:**

- Study information will be communicated to the subjects by the investigator, or designee, and by interactive video.
   After signing the ICF, subjects will be asked to complete a knowledge check (a quiz).
   Subjects will also be shown a list of the ingredients contained in the test products to confirm they have no known allergies or hypersensitivity to any of the ingredients.
- 2. Send study information video (at Screening) and brushing instruction video (at Baseline) to subjects using WeChat.
- 3. Qualifying tactile threshold (g) and Schiff sensitivity scores can be recorded on paper source documents for later transcription into the electronic case report form (eCRF).
- 4. Prior to clinical examinations and assessments, subjects will be shown or reminded how to complete a VAS. Evaporative (air) assessments follow the tactile assessments, with minimum 5 minutes between last tactile assessment and first evaporative (air) assessment (to allow tooth recovery).
  - Visits 1 and 2: maximum force for tactile assessments = 20g
  - Visits 3 and-4: maximum force for tactile assessments = 80g

The clinical examiner should communicate their Schiff sensitivity score to the scribe (non-verbally) before the subject completes the VAS. Examiner and subject should be blinded to each other's scores.

VAS is a qualifying assessment at Baseline ONLY.

5. Test teeth must only be selected from eligible teeth (no dentition exclusions, presence of EAR, MGI = 0 adjacent to the test area only, clinical mobility = 0) with a tactile threshold  $\leq$  20 g and a Schiff sensitivity score  $\geq$  2 at both Screening and Baseline, and VAS  $\geq$  40 mm at Baseline.

Test teeth must have the same Schiff sensitivity score at Screening and Baseline (i.e., Schiff sensitivity score = 2 at Screening and Baseline, or Schiff sensitivity score = 3 at Screening and Baseline)

- 6. Return study supplies to subject after supervised brushing.
- 7. **Subjects randomized to test toothpaste only:** Dispensing staff will show the subject the location of their two test teeth prior to supervised brushing.
- 8. Record AEs from signing of the informed consent form (ICF) until 5 days after last use of study product (or the last study procedure).

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH

Clinical Protocol

Protocol Number: 300026



### 2 INTRODUCTION

Dentine hypersensitivity (DH) has been defined as 'pain derived from exposed dentine in response to chemical, thermal, tactile, or osmotic stimuli which can't be explained as arising from any other dental defect or disease' (Addy, 1985; Canadian Advisory Board on Dentin Hypersensitivity, 2003). The primary aetiological factors associated with the onset of DH include gingival recession and/or enamel loss (e.g., through dental erosion or abrasion), both result in exposure of dentine with patent dentinal tubules (Orchardson, 2000). The hydrodynamic theory of DH hypothesises that an external stimulus (e.g., a temperature/osmotic differential) applied to exposed dentine disrupts the movement of fluid within dentinal tubules (Brännström, 1962). This disruption may stimulate nerve processes in the pulpal area of the dentine including irritation of odontoblasts, pulpal neurons, and even subodontoblastic blood vessels (Hall, 2000), resulting in the characteristic short, sharp pain of DH.

Currently there are two approaches to the management of DH: nerve depolarisation or dentine tubule occlusion. Nerve depolarising agents, typically potassium salts, generally require a period of use (e.g., 14 to 28 days) before their benefit is established. The delivery of potassium ions to the dentine-pulp junction (odontoblastic layer) *via* exposed dentine tubules is believed to result in depolarisation of the afferent nerve membrane thereby interrupting the pain response (Orchardson, 2000). The second approach uses occluding agents which act to physically block or narrow the exposed end of dentinal tubules (by the precipitation of insoluble materials onto the dentine surface and/or within dentinal tubules), thus reducing disruption to dentinal fluid movement in response to an external stimulus (Pashley, 1986).

Stannous fluoride (SnF<sub>2</sub>) has been incorporated into oral hygiene products indicated for the reduction of DH since the 1990s (<u>Schiff, 2006</u>); it provides relief from DH by the occlusion of the dentine tubules through chemical precipitation of stannous oxides and hydroxides. Proctor and Gamble (P&G), Colgate and the sponsor market 0.454% SnF<sub>2</sub> toothpastes indicated for DH relief, with published evidence demonstrating longitudinal clinical efficacy (<u>Ni, 2010</u>; <u>Parkinson, 2011</u>; <u>Makin, 2013</u>).

# 2.1 Study Rationale and Background

The longer-term clinical efficacy of sponsor's 0.454% SnF<sub>2</sub> toothpastes is currently supported by two 8-week DH studies conducted outside China (<u>Parkinson et al, 2013; Parkinson et al, 2015</u>). The Chinese MoH guidelines (<u>Ministry of Health China, 2010</u>) require two clinical studies to support the efficacy of a functional toothpaste, with at least one of these studies (for each claimed benefit) to be conducted in a local Chinese population. Thus, a clinical study in the Chinese population which meets the additional requirements described above is required to support longer-term DH relief claims for the sponsor's 0.454% SnF<sub>2</sub> toothpastes in China.

### 2.2 Benefit/Risk Assessment

Study products are commercially available daily use toothpastes which contain only ingredients with a history of safe use in oral healthcare products. Summary safety information for the acclimatization and study products will be provided on the product labels.

### 2.3 Mechanism of Action/Indication

Occlusion agents act to physically block or narrow dentinal tubules where they open on to the surface of exposed dentine, thereby preventing or reducing disruption to the movement of fluid within the tubule in response to an external stimulus ( $\underline{Addy}$ ,  $\underline{2002}$ ). SnF<sub>2</sub> is one of the most

Clinical Protocol

Protocol Number: 300026



commonly employed tubule-occluding agents included in anti-sensitivity toothpastes. The stannous (tin [II]) ion reacts with water and phosphate minerals found in saliva and dentine tubule fluid to form insoluble deposits (a 'protective' layer) over the surface of the dentine (Parkinson 2011; Parkinson 2013)

# 3 STUDY OBJECTIVES AND ENDPOINTS.

Table 3-1 Study Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary | |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to an evaporative (air) stimulus (as measured by Schiff sensitivity score), compared to a negative control toothpaste, after 12 weeks twice daily use. | Change from Baseline in Schiff sensitivity score at Week 12. |
| Secondary | |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to a tactile stimulus (as measured by tactile threshold), compared to a negative control toothpaste, after 12 weeks twice daily use. | Change from Baseline in tactile threshold (grams [g]) at Week 12. |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to an evaporative (air) stimulus (as measured by Visual Analogue Scale [VAS]), compared to a negative control toothpaste, after 12 weeks twice daily use. | Change from Baseline in VAS (millimeters [mm]) at Week 12. |
| To determine the clinical efficacy of a 0.454% w/w SnF <sub>2</sub> toothpaste in reducing DH to evaporative (air) and tactile stimuli (as measured by Schiff sensitivity score/VAS and tactile threshold, respectively), compared to a negative control toothpaste, after 6 weeks twice daily use. | Change from Baseline in Schiff sensitivity score, tactile threshold (g) and VAS (mm) at Week 6. |
| To determine the clinical efficacy of a 5.0% w/w calcium sodium phosphosilicate (CSPS) toothpaste (positive control) in reducing DH to evaporative (air) and tactile stimuli (as measured by Schiff sensitivity score/VAS and tactile threshold, respectively), compared to a negative control toothpaste, after 6 and 12 weeks twice daily use. | Change from Baseline in Schiff sensitivity score and tactile threshold (g) and VAS (mm) at Week 6 and Week 12. |
| Safety | |
| To evaluate the safety and oral tolerability of the study toothpastes when used twice daily for 12 weeks. | Treatment emergent adverse events (TEAEs) |

The study will be considered successful if the 0.454% SnF<sub>2</sub> toothpaste demonstrates statistically significant, superior anti-hypersensitivity efficacy, compared to negative control, as measured by Schiff sensitivity score at Week 12.

Protocol Number: 300026



### 4 STUDY DESIGN

### 4.1 **Overall Design**

This will be a single centre, 12-week, randomised, controlled, examiner-blind, 3-treatment arm, parallel group design, stratified (by maximum Baseline Schiff sensitivity score of the 2 selected test teeth) clinical study investigating the clinical efficacy of a 0.454% SnF<sub>2</sub> toothpaste for the relief of DH in a Chinese population. A 5.0% CSPS toothpaste with clinically proven longerterm DH efficacy in the Chinese population will be included in the study as a positive control. The clinical efficacy of both anti-sensitivity toothpastes will be compared with that of a regular fluoride toothpaste (negative control), with no known anti-sensitivity properties.

Two stimuli will be employed to evaluate the DH efficacy of the test toothpaste. A tactile stimulus will be administered using a constant pressure probe (Yeaple Probe (Polson, 1980)); subject response to the stimulus determines the tactile threshold in grams (g). An evaporative (air) stimulus will be administered using a dental air syringe; subject response to the stimulus will be evaluated by a dental examiner using the Schiff sensitivity scale (Schiff, 1994) and a subject-completed VAS (mm). DH will be assessed at Screening, Baseline (Day 1), Week 6 and Week 12.

- At Screening, tactile sensitivity will be assessed for all eligible teeth identified by oral **examination** (i.e. no dentition exclusions, presence of EAR, MGI = 0 adjacent to the test area only, clinical mobility = 0), followed by evaporative (air) sensitivity (with Schiff sensitivity score and VAS) for eligible teeth with tactile threshold  $\leq 20g$ .
- At Baseline, tactile sensitivity will be assessed for all eligible teeth identified at **Screening** (i.e. no dentition exclusions, presence of EAR, MGI = 0 adjacent to the test area only, clinical mobility = 0, tactile threshold  $\leq$  20g at Screening, Schiff sensitivity score  $\geq 2$  at Screening); followed by evaporative (air) sensitivity (with Schiff sensitivity score and VAS) for all eligible teeth identified at Screening with Baseline tactile threshold  $\leq 20g$ .

On completion of the Baseline assessments, two test teeth will be selected for continued assessment of tactile and evaporative (air) sensitivity at subsequent visits. Each test tooth must comply with the following selection criteria:

- No dentition exclusions, presence of EAR, MGI = 0 adjacent to the test area only and clinical mobility = 0
- Tactile threshold  $\leq 20g$  at Screening and Baseline
- Schiff sensitivity score  $\geq 2$  at Screening and Baseline
- VAS  $\geq$  40 mm at Baseline only
- Test teeth must have the <u>same</u> Schiff sensitivity score at Screening <u>and</u> Baseline Schiff sensitivity score = 2 at Screening and Baseline, OR Schiff sensitivity score = 3 at Screening and Baseline

Qualifying subjects will be stratified according to the maximum Baseline Schiff sensitivity score of their two test teeth and randomised to one of the 3 study toothpastes. Randomised subjects will brush their teeth twice daily (morning and evening) with their assigned study toothpaste for the duration of the 12-week treatment period.

Safety and oral tolerability of the study products will be monitored throughout the study by review of subject- and examiner-reported AEs.

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH

Clinical Protocol

Protocol Number: 300026



# 4.2 Scientific Rationale for Study Design

A randomised, controlled, examiner-blind, parallel group design is a recognised approach for investigating the clinical efficacy of a product for the relief of DH (Holland, 1997).

The longer-term clinical efficacy of the sponsor's 0.454% SnF<sub>2</sub> toothpastes is currently supported by two 8-week DH studies conducted outside China (Parkinson et al, 2013; Parkinson et al, 2015). Longer-term DH studies evaluating an alternative occlusion technology (CSPS) in China employed a longer treatment period (Hall et al, 2017 11 weeks; In order to establish longitudinal performance for the test toothpaste, with greater opportunity for its clinical benefits to be observed, a 12 week treatment period will be employed here (Murray, 1994; Irwin, 1997). To comply with Chinese MoH guidelines for the testing of functional (desensitising) toothpastes, a single interim assessment timepoint will be included after 6 weeks' treatment ('Sensitivity levels are to be examined and recorded at the baseline, mid-trial and end-trial stages'; Ministry of Health (China), 2010).

In line with published recommendations for the design and conduct of DH studies (Holland, 1997) and the requirements of the Chinese MoH guidelines for the testing of functional (desensitising) toothpastes (Ministry of Health (China), 2010), two independent stimuli will be employed (tactile and thermal (evaporative air) stimuli) to evaluate the efficacy of the 0.454% SnF<sub>2</sub> toothpaste. To avoid inter-assessor variability, the same clinical examiner should be responsible for the administration of a given stimulus (tactile or evaporative (air)) and the conduct of the associated examiner-assessed DH measure from Screening until the end of the study. DH will be assessed at Screening, Baseline (pre-treatment) and following 6 and 12 weeks of treatment.

The age range over which an individual can experience DH is wide (early teens to 70s) (Fischer et al, 1992), with peak incidence known to occur between the ages of 20-40 years (Flynn et al, 1985). The fall in prevalence observed in later decades reflects age-related changes in the dentine and pulp of the tooth which act to reduce both dentine permeability and the tooth's response to external triggers of DH (Pashley, 2008; Seltzer and Bender, 1975). The dental pain experienced by much older members of the population is less likely to be diagnosed as DH (Rees, 2000), thus an age range of 18-70 years has been selected for this study to target individuals with tooth sensitivity due to DH.

While there is no published evidence to indicate that gender impacts the pathophysiology of DH, a national DH survey conducted in rural China in 2009 reported a greater proportion of females with DH compared to males (female 35.8%; male 23.4%) (Liang, 2017). To ensure the current study population is representative of the Chinese population being studied, the study site will aim to recruit a female:male ratio of approximately 3:2.

According to ICH guidelines (ICH E6 (R2) Good clinical practice | European Medicines Agency (europa.eu), for a study to be classed as double blind, the subject, investigator, clinical examiners, monitors, data analysts, and staff involved in determining subject eligibility/ assessing compliance should be blinded to the treatment a subject receives. However, given it will not be possible to ensure identical appearance, flavour and packaging for the three commercial toothpastes to be evaluated in this study, the study is described as 'examiner blind'.

In line with the Chinese MOH guidelines (Ministry of Health (China), 2010) for the testing of functional (desensitising) toothpastes, a regular fluoride toothpaste with no known (or claimed) anti-sensitivity efficacy will be included as the negative control (Crest Cavity Protection Fresh Lime; China commercial product). In addition, a 5.0% CSPS toothpaste (Sensodyne Repair & Protect; China commercial product) with proven DH efficacy in the Chinese population (in

Clinical Protocol

Protocol Number: 300026



clinical studies that satisfied current (at time of writing) Chinese MoH guidelines: sponsor clinical studies Hall et al, 2017 and will be included in the study as a positive control (i.e., as a benchmark of performance in the Chinese population for 'study validation'). Given the primary objective is to demonstrate statistical superiority for the test toothpaste compared to negative control in change from Baseline in Schiff sensitivity score at Week 12, qualifying subjects will be randomised to study treatment using a 2:2:1 allocation ratio (Test: Negative Control: Positive Control).

Subjects using anti-sensitivity products as part of their normal oral hygiene routine will be excluded (their own oral hygiene products will be checked for presence of known anti-sensitivity ingredients at Screening); if they are continuing to experience DH, they are unlikely to respond to use of a sensitivity toothpaste in the current study.

Subjects will be asked to describe their typical daily oral care regimen at Screening. To help maintain study product in the oral cavity for the duration of each timed brushing, any subject who habitually rinses with water during toothbrushing (self-reported) will be excluded from the study. Similarly, at Baseline, following review of the brushing videos, any subjects who rinsed during brushing with the acclimatisation toothpaste will be excluded.

Clinical trials evaluating pain-related end points can be prone to 'placebo effects' (Addy, 1985; West, 1997); such effects are frequently observed in DH studies. A study conducted to evaluate the natural history of the DH condition also highlighted the existence of a 'no treatment' effect, characterised by an improvement in sensitivity simply as a result of study participation (Leight, 2008). Analyses of sponsor data from earlier DH efficacy studies indicate (i) subjects with a lower frequency of DH symptoms may exhibit greater 'placebo'/ 'no treatment' effects (sponsor clinical study: 216953) and (ii) subjects with different qualifying Schiff sensitivity scores at Screening and Baseline for one or both test teeth may also exhibit greater 'placebo'/ 'no treatment' effects (sponsor clinical study: 216954).

To help minimise the potential impact of such effects:

- An acclimatisation period (2-4 weeks) will precede the Baseline visits. During this period, study subjects will brush twice daily with the regular fluoride toothpaste and toothbrush provided (in place of their normal oral hygiene products) and record each timed brushing occasion in a diary. The acclimatisation period will also help standardise oral hygiene practice across the study population prior to treatment.
- Subjects will complete a Screening Questionnaire (<u>Appendix 15.2</u>) at Visit 1; those who report experiencing DH symptoms only 'several times a month', 'once a month' or 'less than once a month' will be excluded from the study.
- Each selected test tooth must have the same qualifying Schiff sensitivity score at the Screening <u>and</u> Baseline visits (i.e., Schiff sensitivity score = 2 at Screening <u>and</u> Baseline, or Schiff sensitivity score = 3 at Screening and Baseline).

On completion of the Baseline assessments, the clinical examiner will select two test teeth from those that qualified at Screening (Visit 1) and Baseline (Visit 2) for assessment of tactile and evaporative (air) sensitivity at all subsequent visits (<u>Table 4-1</u>). The selection of two 'test teeth' to evaluate changes in DH is common practice in sensitivity studies (<u>Schiff, 1994</u>). Qualifying subjects will be stratified according to the maximum Schiff sensitivity score of their two selected test teeth to ensure treatment groups are balanced for DH severity.

DH is an episodic condition; symptoms are known to vary spontaneously (West, 2008, West et al., 2013). Baseline clinical values that would support enrolment may represent random highs

Clinical Protocol

Protocol Number: 300026



that could be followed by regression to the mean, leaving the subject or selected test tooth without the condition under investigation during the treatment period. To help minimise the potential for this to occur on the current study, randomised subjects will be required to demonstrate consistency in DH response at both the Screening and Baseline visits.

- Randomised subjects must have a minimum of two eligible teeth (no dentition exclusions, presence of EAR, MGI = 0 adjacent to the test area only, clinical mobility = 0) with a tactile threshold ≤ 20 g and a Schiff sensitivity score ≥ 2 at both Screening and Baseline.
- Test teeth can only be selected from eligible teeth identified at Screening (no dentition exclusions, presence of EAR, MGI = 0 adjacent to the test area only, clinical mobility = 0), with a tactile threshold ≤ 20 g and a Schiff sensitivity score ≥ 2 at both Screening and Baseline and with VAS ≥ 40 mm at Baseline only.
- Test teeth must have the same Schiff sensitivity score at Screening and Baseline.

Table 4-1 Eligibility Checks for Test Tooth Selection

| Screening Assessments (Visit 1) | | | | | Baseline Assessments (Visit 2) | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Dentition<br>Exclusions | EAR | MGI* | Clinical<br>Mobility | Tactile<br>Threshold | Schiff<br>Sensitivity<br>Score | Eligible<br>Tooth | Tactile<br>Threshold | Schiff<br>Sensitivity<br>Score | VAS | Test<br>Tooth |
| None | Yes | 0 | 0 | $\leq$ 20g | 2 | Yes | $\leq$ 20g | 2 | ≥ 40mm | Yes |
| None | Yes | 0 | 0 | ≤20g | 3 | Yes | ≤ 20g | 3 | ≥ 40mm | Yes |
| None | Yes | 0 | 0 | ≤ 20g | 2 | Yes | ≤ 20g | 3 | ≥ 40mm | No |
| None | Yes | 0 | 0 | ≤20g | 3 | Yes | ≤20g | 2 | ≥ 40mm | No |

Eligibility against each selection criterion is determined sequentially.

VAS is completed at Screening <u>and</u> Baseline, but is a qualifying measure for Test Tooth Selection at Baseline **ONLY**.

### 4.3 Justification for Dose

Study products are toothpastes, intended for topical oral use, and will be applied by toothbrushing using a manual toothbrush.

The usage regimen of twice daily brushing (morning and evening) will be the same for all subjects, based on widely recommended oral hygiene practice and typical consumer habit. Study subjects will brush for 1-timed minute with their assigned study toothpaste on each brushing occasion in line with typical brushing times specified for similar DH efficacy studies (Parkinson, 2011; Makin, 2013; Hall et al., 2017; Docimo et al., 2009). Subjects allocated to the test toothpaste will be instructed to brush their two test teeth first, to ensure their sensitive teeth are treated, then their whole mouth for 1-timed minute. The usage regimen specified for the negative and positive control products is aligned with the usage instructions provided on the commercial packaging of both toothpastes.

After 12 weeks ( $85 \pm 4$  days) twice daily usage, each subject should complete between 162-178 brushings with their randomized product. Subjects will complete a supervised brushing with their assigned study toothpaste at the end of each study visit (while still at the study site) to

<sup>\*</sup>Adjacent to the test area only

Clinical Protocol

Protocol Number: 300026



enable staff to confirm correct usage and to encourage compliance with the required usage regimen for the duration of the study.

Tongue cleaning forms an integral part of typical oral hygiene practice for many Chinese consumers; it will be permitted during the current study (using the toothbrush provided), after completing each 1-minute toothbrushing with study toothpaste but before the 10ml water rinse. Tongue brushing is not permitted while toothbrushing.

To help ensure the study toothpaste is retained in the oral cavity for the 1-minute brushing time, subjects must not rinse with water or expectorate during toothbrushing.

A recent consumer study (sponsor data on file) observed rinsing with variable, often copious amounts of water following toothbrushing to be common practice in Chinese consumers. To standardise rinsing practice across the study population, all subjects will be instructed to rinse once with water (10 ml dispensed from a dosing cup) after each brushing occasion.

# 4.4 End of Study Definition

A subject will be considered to have completed the study if they have completed all phases of the study including the last visit or the last scheduled procedure shown in the Schedule of Activities.

The end of this study is defined as the date of the last scheduled procedure, as described in the Schedule of Activities (<u>Table 1-1</u>), for the last subject.

# 5 STUDY POPULATION

# 5.1 Type and Planned Number of Subjects

The study will be conducted in a Chinese population (in China). Subjects will be male or female, with a minimum of 20 natural teeth, a self-reported history of tooth sensitivity and at least two teeth with clinical examiner-confirmed DH (tactile threshold  $\leq 20$  g and Schiff sensitivity score  $\geq 2$  at both Screening and Baseline; VAS  $\geq 40$  mm at Baseline). In addition, the selected test teeth must demonstrate a consistent response to the evaporative (air) stimulus at the Screening and Baseline visits (Schiff sensitivity score = 2 at Screening and Baseline, or Schiff sensitivity score = 3 at Screening and Baseline).

Sufficient subjects will be screened to randomize approximately 240 subjects to study treatment to ensure approximately 235 subjects complete the study (approximately 94 each for test toothpaste and negative control, and 47 for positive control), allowing for approximately 2% dropouts after randomization, as observed in previous clinical studies conducted in China.

Whilst the study products are not contra-indicated for pregnancy and breastfeeding, pregnant and/or lactating females will be excluded from this study due to the increased prevalence and severity of gingivitis and periodontal disease observed during pregnancy (Samant et al., 1976) and breastfeeding (Aghazadeh et al., 2019) which, together with the increased amounts of calculus and plaque observed during pregnancy, could impact DH assessments (Samant et al., 1976).

An enrolled subject is one who has agreed to participate in the clinical study following completion of the informed consent process (directly or via their legally authorized representative) and successfully met the eligibility criteria to proceed beyond the screening visit as described in the protocol design.

Clinical Protocol

Protocol Number: 300026



This study can fulfill its objectives only if appropriate subjects are enrolled. The following eligibility criteria are designed to select subjects for whom participation in the study is considered appropriate. All relevant medical and non-medical conditions should be taken into consideration when deciding whether a subject is suitable for this protocol.

Subject eligibility to participate in the clinical study should be reviewed and documented by an appropriate member of the investigator study team before a subject is included in the study.

### 5.2 Inclusion Criteria

An individual must meet all of the following inclusion criteria to be eligible for enrollment into the study:

- 1. Provision of a signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study before any study procedures are performed.
- 2. Male or female who, at the time of screening, is between the ages of 18 to 70 years inclusive.
- 3. Subject who is willing and able to understand and comply with scheduled visits, product usage requirements and other study procedures.
- 4. Subject in good general, oral and mental health with, in the opinion of the investigator or medically qualified designee, no clinically significant or relevant abnormalities in medical history, or upon oral examination, that would impact the subject's safety or wellbeing, or the outcomes of the study, if they were to participate in the study, or affect the subject's ability to understand and follow study procedures and requirements.
- 5. Subject who owns a smartphone with WeChat application installed.

# 6. At Screening (Visit 1)

Subject must have:

- a) Self-reported history of tooth sensitivity lasting more than 6 months but not more than 10 years and experience DH symptoms at least 'once a week' or more frequently (Screening Questionnaire, <u>Appendix 15.2</u>).
- b) Good general oral health, with a minimum of 20 natural teeth.
- c) Minimum of **two** accessible, non-adjacent teeth (incisors, canines, pre-molars), preferably in different quadrants, with clinically confirmed DH.

Each eligible tooth must meet <u>all</u> the following criteria:

- i. Exposed dentine due to facial/cervical erosion, abrasion or gingival recession (EAR).
- ii. MGI = 0 directly adjacent to the exposed dentine (i.e., the test area) only.
- iii. Clinical mobility = 0.
- iv. DH as evidenced by qualifying levels of tactile and evaporative (air) sensitivity (tactile threshold  $\leq 20g$  and Schiff sensitivity score  $\geq 2$ ).

Clinical Protocol

Protocol Number: 300026



### 7. At Baseline (Visit 2):

All teeth identified at Screening (Visit 1) as eligible for Baseline assessments will be reassessed for tactile sensitivity first; eligible teeth with Baseline tactile threshold  $\leq 20$ g will then be re-assessed for evaporative (air) sensitivity.

Subjects must have:

A minimum of two non-adjacent, accessible teeth (incisors, canines, pre-molars), preferably in different quadrants, with clinically confirmed DH as evidenced by qualifying levels of tactile and evaporative (air) sensitivity:

- a) Tactile threshold  $\leq 20g$  at Screening and Baseline
- b) Schiff sensitivity score  $\geq 2$  at Screening and Baseline.
- c)  $VAS \ge 40$  mm at Baseline.

The clinical examiner will select <u>two</u> 'test teeth' from those eligible teeth which meet the tactile threshold <u>and</u> Schiff sensitivity score criteria at both Screening <u>and</u> Baseline, and the VAS criterion at Baseline.

Each test tooth must demonstrate a consistent DH response to the evaporative (air) stimulus at both Screening and Baseline:

| 8 |
|---|
| <b>Screening</b> Schiff sensitivity score = 2 <u>and</u> <b>Baseline</b> Schiff sensitivity score = 2 |
| OR |
| <b>Screening</b> Schiff sensitivity score = 3 <u>and</u> <b>Baseline</b> Schiff sensitivity score = 3 |

The procedure for selecting test teeth is summarised in **Table 4-1**.

### 5.3 Exclusion Criteria

An individual who meets any of the following exclusion criteria will be excluded from the study:

- 1. Subject who is an employee of the study site, either directly involved in the conduct of the study or a member of their immediate family; or an employee of the study site otherwise supervised by the investigator; or a sponsor employee directly involved in the conduct of the study or a member of their immediate family.
- 2. Subject who is participating in, or has participated in, other studies (including non-medicinal studies) involving investigational product(s) within 30 days of Screening (Visit 1).
- 3. Subject who is participating in, has participated in, a study evaluating a tooth desensitising treatment within 8 weeks of Screening (Visit 1).
- 4. Subject who is using, or has used, an oral care product indicated for DH relief within 8 weeks of Screening (Visit 1). Subjects will be required to bring their current oral care products to Visit 1 for staff to verify the absence of known anti-sensitivity ingredients and DH claims.
- 5. Subject who has had a professional de-sensitising treatment within 8 weeks of Screening (Visit 1).
- 6. Subject who habitually rinses with water during toothbrushing (self-reported at Screening (Visit 1)).
- 7. Subject seen to rinse with water while brushing with the acclimatization toothpaste during

Clinical Protocol

Protocol Number: 300026



review of their brushing compliance videos at Baseline (Visit 2).

- 8. Subject with known or suspected intolerance or hypersensitivity to the study products or any of their stated ingredients (or closely related compounds).
- 9. Subject who is unwilling or unable to comply with product usage instructions (Section 4.3) or Lifestyle Considerations (Section 5.5) as described in the protocol.
- 10. Female subject who is pregnant or intending to become pregnant during the study (self-reported).
- 11. Female subject who is breastfeeding.
- 12. Subject with a recent history (within the last year) of alcohol and/or substance abuse.
- 13. Subject with, in the opinion of the investigator or medically qualified designee, an acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study product administration or may interfere with the interpretation of study results and, in the judgment of the investigator or medically qualified designee, would make the subject inappropriate for entry into this study.
- 14. Subject taking daily doses of medications or traditional herbal treatments which, in the opinion of the investigator or medically qualified designee, could interfere with their perception of pain.
  - Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilisers, anti-depressants, moodaltering and anti-inflammatory drugs.
  - Examples of herbal treatments include clove oil, olive oil or other treatments directly applied to the oral cavity for the treatment of oral health conditions.
- 15. Subject taking daily doses of a medication which, in the opinion of the investigator or medically qualified designee, is causing xerostomia.
- 16. Subject who requires antibiotic prophylaxis for dental procedures.

# 17. At Screening (Visit 1)

Subject who has taken antibiotics within 2 weeks of their Screening visit.

### 18. At Baseline (Visit 2)

Subject who has taken antibiotics within 2 weeks of their Baseline visit (during the acclimatisation period).

- 19. Subject who has had a professional or self-applied tooth bleaching procedure within 8 weeks of Screening (Visit 1).
- 20. Subject who has had dental prophylaxis within 4 weeks of Screening (Visit 1).
- 21. Subject who has had treatment for periodontal disease (including surgery) within 12 months of Screening (Visit 1).
- 22. Subject who has had scaling or root planning within 3 months of Screening (Visit 1).
- 23. Subject with a tongue or lip piercing.
- 24. Subject with, in the opinion of the investigator or medically qualified designee, gross periodontal disease.

Clinical Protocol

Protocol Number: 300026



- 25. Subject with evidence of gross intra-oral neglect or the need for extensive dental therapy.
- 26. Subject with a fixed or removable partial prosthesis which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
- 27. Subject with multiple dental implants which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
- 28. Subject with fixed or removable orthodontic braces/bands or a fixed orthodontic retainer.

### 29. SPECIFIC DENTITION EXCLUSIONS FOR 'TEST TEETH':

- a) Tooth with evidence of current or recent caries or reported treatment of decay within 12 months of Screening (Visit 1).
- b) Tooth with exposed dentin but with deep, defective or facial restorations.
- c) Tooth with full crown or veneer.
- d) Tooth adjacent to a bridge abutment or crown which, in the opinion of the investigator or medically qualified designee, would impact study outcomes.
- e) Sensitive tooth with contributing aetiologies other than erosion, abrasion or recession to exposed dentine.
- f) Sensitive tooth, in the opinion of the investigator or medically qualified designee, not expected to respond to treatment with an anti-sensitivity toothpaste.
- 30. Subject who has previously been enrolled in this study.
- 31. Any subject who, in the opinion of the investigator or medically qualified designee, should not participate in the study.

### 5.4 Randomization Criteria

Subjects who satisfy all selection criteria will be randomized into the study. Randomisation numbers will be assigned in ascending numerical order as each subject is determined to be fully eligible.

Subjects will be stratified by the maximum Baseline Schiff sensitivity score of their two selected test teeth. The stratification factor will give rise to two strata.

- **Stratum 1:** Maximum Schiff sensitivity score = 2
- **Stratum 2:** Maximum Schiff sensitivity score = 3

Within each stratum, subjects will be randomized to test toothpaste, negative control or positive control with 2:2:1 allocation ratio using permuted randomised blocks (see Section 12.1).

# 5.5 Lifestyle Considerations

If, in the opinion of the investigator or medically qualified designee, a subject has not complied with a study restriction (oral hygiene, dietary or alcohol-related) prior to a study visit or cannot attend a study visit, every effort will be made to reappoint them within the permitted visit tolerances (see Schedule of Activities, <u>Table 1-1</u>). The reason for re-appointment will be documented in the electronic case report form (eCRF).

Clinical Protocol

Protocol Number: 300026



If re-appointment is not possible, the following visit specific actions should be taken:

- **Baseline (Visit 2):** if the subject cannot be reappointed (within the 2-4 week visit tolerance), they will be withdrawn from the study. No clinical efficacy assessments will be performed. The subject may be replaced.
- Week 6 (Visit 3): if the subject cannot be reappointed (within the visit tolerance) the subject will continue in the study. No clinical efficacy assessments will be performed.
- Week 12 (Visit 4): if the subject cannot be reappointed (within the visit tolerance), they will be withdrawn from the study. No clinical efficacy assessments will be performed. The subject will not be replaced.

### 5.5.1 Oral Care Restrictions

# For the Duration of the Study: From Screening (Visit 1) to the Subject's Last Study Visit

- Subjects should stop using their own oral care products
- Subjects should not use any other oral care products (e.g., toothpastes, toothbrushes, oral rinses, tongue cleaners, whitening/bleaching products, interdental cleaning products) than those provided during the study.

Note: Dental floss can be used but only to remove impacted food.

• Subjects should not chew gum.

### Before a Clinical Assessment Visit: Baseline (Visit 2), Week 6 (Visit 3), Week 12 (Visit 4)

• Subjects will refrain from all oral hygiene procedures for at least 8 hours prior to their appointment (subjects will be sent a WeChat reminder the day before their appointment to remind them of this).

### 5.5.2 Dietary and Alcohol Restrictions

### Before a Clinical Assessment Visit: Baseline (Visit 2), Week 6 (Visit 3), Week 12 (Visit 4)

- Subjects must not eat or drink for at least 2 hours before a clinical assessment visit.
  - **Note:** Small sips of room-temperature water are permitted to take medications or to relieve a dry mouth up to 1 hour before their appointment time
- Subjects should refrain from excessive alcohol consumption for 24 hours before a clinical assessment visit.

### 5.5.3 Covid-19

Local Chinese guidelines and/or clinical site requirements will be followed.

### 5.5.4 Contraception

Given the study products are commercially available toothpastes, regulated as General Goods in China, and no drugs will be utilised in this clinical study, pregnancy testing and contraceptive requirements are not deemed necessary.

Protocol Number: 300026



### 5.6 Screen Failures

Screen failures are defined as subjects who consent to participate in the clinical study but are not subsequently randomised. To ensure transparent reporting of screen failure subjects, a minimal set of screen failure information will include demography, screen failure details (e.g., withdrawal of consent), eligibility criteria, any protocol deviations and any AEs, as applicable.

Individuals who do not meet the criteria for participation in this study (screen failure) may not be re-screened.

# 5.7 Sponsor's Qualified Medical Personnel

Contact information for the sponsor's appropriately qualified and experienced medical/dental personnel or Clinical Research Scientist (CRS) for the study is documented in the Study Contact List located in the investigator site master file held at the study site.

The contact number is only to be used by study staff seeking advice on medical/dental questions or problems in the event that the established communication pathways between the study site and the sponsor's study team are not available.

The contact number is not intended for direct use by study subjects. To facilitate access to appropriately qualified sponsor personnel on study-related medical/dental questions or problems, subjects will be provided with a contact card. The contact card will provide, as a minimum, protocol identifiers, the subject's study identification number, contact information for the study site, and contact details in the event that the study site cannot be reached to provide advice on a medical question or problem identified by a healthcare professional other than the investigator.

### 5.8 Clinical Assessor Qualifications

The examiners responsible for the clinical efficacy measures will be qualified dentists, trained in the clinical assessment of DH (tactile and evaporative (air) sensitivity).

Additional qualified dentists, not trained in the clinical assessment of DH, will be permitted to conduct the oral (OST/OHT) examinations required at each study visit.

Protocol Number: 300026



### 6 STUDY PRODUCTS

For the purposes of this study, per International Conference on Harmonization (ICH) guidelines, and sponsor policy, study intervention is defined as any investigational intervention(s), marketed product(s), placebo, or medical device(s) intended to be administered to a study participant according to the study protocol.

# 6.1 Study Product Supplies

The following study products will be supplied by the sponsor's Clinical Supplies Department:

Table 6-1 Study Product Supplies

| Product<br>Description | Test Toothpaste | Reference<br>Toothpaste<br>(Positive Control) | Reference Toothpaste<br>(Negative Control) |
|---|---|---|---|
| Product<br>Name** | 0.454% w/w SnF <sub>2</sub> toothpaste (Sensodyne Sensitivity & Gum*) | 5.0% w/w CSPS<br>toothpaste<br>(Sensodyne Repair &<br>Protect*) | Regular Fluoride<br>toothpaste<br>(Crest Cavity Protection<br>Fresh Lime*) |
| Fluoride<br>Content | 1100 ppm fluoride as SnF <sub>2</sub> | 1150 ppm fluoride as<br>NaF | 1150 ppm ppm<br>fluoride as NaF |
| MFC | CCI | CCI | N/A |
| Pack Design | One carton containing 6 over-wrapped tubes of toothpaste | | |
| Dispensing<br>Details | Baseline (Visit 2): One carton | | |
| Product<br>Application | Dose the toothbrush with a strip of toothpaste (a ribbon of toothpaste across the full brush head) on each brushing occasion | | |
| Route of Administration | Topical Oral Use | | |
| Usage<br>Instructions <sup>†</sup> | Brush the two test teeth first, then the whole mouth (all teeth) for 1-timed minute, twice daily (morning and evening). After brushing, rinse once with 10 ml water using the measuring cup provided. | Brush the whole mouth (all teeth) for 1-timed minute. After brushing, rinse once with 10 ml water using the measuring cup provided. | |
| Return<br>Requirements | All used/un | all used/unused samples to be returned | |

<sup>\*</sup>Chinese commercial product

<sup>†</sup> After completing each toothbrushing, subjects will be permitted to clean their tongue using the toothbrush provided (but this is not a study requirement). Tongue brushing must be completed after toothbrushing but before rinsing with 10 ml water.

Clinical Protocol

Protocol Number: 300026



### Table 6-2 Acclimatization Product

| <b>Product Description</b> | Acclimatization Toothpaste |
|---|---|
| Product Name | Regular fluoride toothpaste (Crest Cavity Protection Fresh Lime*) |
| Fluoride Content | 1150ppm ppm fluoride as NaF |
| MFC | N/A |
| Pack Design | One carton containing 2 over-wrapped tubes of toothpaste |
| <b>Dispensing Details</b> | Screening (Visit 1): One carton |
| <b>Product Application</b> | Dose the toothbrush with a strip of toothpaste (a ribbon of toothpaste across the full brush head) on each brushing occasion |
| Route of Administration | Topical Oral Use |
| Usage Instructions† | Brush the whole mouth (all teeth) for 1-timed minute. After brushing, rinse once with 10 ml water using the measuring cup provided. |
| Return Requirements | All used/unused samples to be returned |

<sup>\*</sup>Chinese commercial product

# Table 6-3 Sundry Items

Sundry Items to be supplied:

| | Cumplied | Pack Design | | Return/Disposal Details | |
|---|---|---|---|---|---|
| Item | Supplied<br>By | | Dispensing Details | Used<br>Samples | Unused<br>Samples |
| Lion Thin<br>Bristle | | Commercial pack | Screening (Visit 1): One toothbrush | Destroy at site | Return to sponsor |
| toothbrush (Chinese | | | Baseline (Visit 2): One toothbrush | using site<br>disposal | |
| commercial product) | | | Week 6 (Visit 3): One toothbrush | procedures | |
| Countdown timer | Sponsor or designated | Commercial pack containing 1 timer | Screening (Visit 1) | | |
| Measuring | vendor | N/A | Screening (Visit 1): 4 cups | Subject to keep | |
| cups | | | Baseline (Visit 2): 12 cups | or destroy at site using site disposal | |
| Opaque | | 27/4 | Screening (Visit 1): One bag | procedures | |
| plastic bags | | N/A | Baseline (Visit 2): One bag | | |

<sup>†</sup> On completing each toothbrushing, subjects will be permitted to clean their tongue using the toothbrush provided (but this is not a study requirement). Tongue brushing must be completed after toothbrushing but before rinsing with 10 ml water.

Clinical Protocol

Protocol Number: 300026



For further information, please refer to the Global Clinical Supplies Packaging and Labelling Proposal. The sponsor will ensure copies of the diary (including toothpaste usage instructions), clinical assessment score sheets and Subject Contact Cards are provided to the study site.

Detailed instructions for the return of study supplies for accountability checks and subsequent destruction which will be provided by the sponsor during the study in time for study close out.

### 6.1.1 Dosage Form and Packaging

All study products (test, negative control, positive control and acclimatization products) are toothpastes, intended for topical oral use, and will be applied using a manual toothbrush. All will be sourced in China.

All toothpastes will be provided to the clinical study site in their commercial packs, overwrapped in white vinyl (to mask their identity and obscure any branding) with a study label affixed. The content of the product labels will be in accordance with all applicable regulatory requirements and will be the responsibility of the sponsor's Global Clinical Supplies Department. Each study label will contain, but not be limited to, protocol number, directions for use and storage requirements.

Each subject will receive sufficient tubes of the acclimatization toothpaste and their assigned study toothpaste to cover usage during the acclimatization and treatment periods, respectively. Sundry items will be supplied in their commercial packaging for dispensing by study staff as required.

Care should be taken with the supplied products and their labels to ensure they are maintained in good condition. It is important that all labels remain intact and legible for the duration of the study. Subjects should be instructed to not remove or deface any part of the over-wrapping or study label.

All products supplied are for use only in this clinical study and should not be used for any other purpose.

### 6.1.2 Product Dispensing

Subjects will be assigned to study product in accordance with the randomization schedule generated by a sponsor-approved vendor, prior to the start of the study, using validated software.

The product dispensing area will be separate from the clinical examination area. Study toothpastes will be dispensed per protocol in blinded fashion to the subject, by trained study personnel. These staff members will not be involved in any safety or clinical efficacy assessments or any other aspect of the study that could be influenced by knowing which product a subject has been assigned to. An additional member of the study staff will verify the dispensing procedure has been completed accurately for each subject.

A record of product dispensing to each subject will be maintained in the dispensing log; completion of the dispensing procedure will be recorded in the eCRF.

### 6.2 Administration

Subjects will self-administer the acclimatization toothpaste (from Visit 1 to Visit 2) and their assigned study toothpaste (from Visit 2 to Visit 4) according to the usage instructions provided by study personnel at the study site and record each brushing in their diary.

Clinical Protocol

Protocol Number: 300026



To help ensure subjects fully understand the amount of toothpaste to use, the brushing instructions and how to complete the diary:

- Screening (Visit 1): Staff will demonstrate dispensing a full ribbon of toothpaste along the length of the toothbrush head to each qualifying subject and supervise their first brushing with the acclimatization toothpaste/diary completion at the end of the visit, after all clinical assessments have been completed.
- **Baseline (Visit 2):** Staff will check the dispensing of a full ribbon of toothpaste by each randomized subject and supervise the first brushing with their assigned study toothpaste/diary completion. Staff will clearly show subjects randomized to test toothpaste the location of their 2 test teeth prior to starting their supervised brushing.
- Week 6 (Visit 3): Staff will supervise each subject brushing with their assigned study toothpaste/completing their diary at the end of the visit, after all clinical assessments have been completed.

On-site administration of study products will be recorded in the dispensing log and the eCRF.

# 6.2.1 Product Dosing Errors

In this study, dosing errors may result from the administration or consumption of the wrong product, by the wrong subject, in the wrong way. Such dosing errors should be captured in the eCRF. Dosing errors are reportable irrespective of the presence of an associated AE, including:

- Dosing errors involving subject exposure to any of the study products.
- Potential dosing errors or uses outside of what was foreseen in the protocol that do or do not involve the participating subject.

If a dosing error is accompanied by an AE, as determined by the investigator or medically qualified designee, the dosing error and any associated AEs are to be captured in the eCRF AE form.

### 6.2.2 Overdose

An overdose is a deliberate or inadvertent administration of a product at an amount higher than specified in the protocol. Overdose is not likely to occur in this study.

Overdose per se is not an AE. However, any clinical sequelae of an overdose should be reported as an AE (and serious adverse event [SAE], if appropriate). For reporting, follow the AE and SAE reporting instructions.

# 6.3 Study Product Storage

The investigator or designee must confirm appropriate temperature conditions have been maintained during transit for all study products received and any discrepancies are reported and resolved before use according to the supplied shipping documentation.

The investigator, or designee, will ensure that all study products are stored in a secured area with controlled access under required storage conditions and in accordance with applicable regulatory requirements and the product labels.

Site systems must be capable of measuring and documenting (e.g., via a log), at a minimum, the daily minimum and maximum temperatures for all site storage locations, as applicable (including frozen, refrigerated, and/or room-temperature products). This should be captured

Clinical Protocol

Protocol Number: 300026



from the time of first product receipt throughout the study. Even for continuous monitoring systems, a log or site procedure that ensures active daily evaluation for excursions should be available. The operation of the temperature-monitoring device/storage unit (e.g., refrigerator), as applicable, should be regularly inspected to ensure it is maintained in working order.

Any excursions from the product-label storage conditions should be reported to appropriate site staff upon discovery and communicated to sponsor as soon as possible. The site should actively pursue options for returning the product to the storage conditions as described in the labeling, as soon as possible. Excursions from the storage requirements, including any actions taken, must be documented as a protocol deviation and reported to the Sponsor.

Once an excursion is identified, the affected product (or products) must be quarantined and not used until the sponsor provides documentation of permission to use. Use of any of the affected product(s) prior to sponsor approval will be considered a protocol deviation.

Site staff will instruct subjects on the proper storage requirements for all take-home products.

# 6.4 Study Product Accountability

All products supplied are for use only in this clinical study and should not be used for any other purpose.

All study products must be received by a designated person at the study sites, handled and stored safely and properly, and kept in a secured location to which only the staff have access. Upon receipt, all study products should be stored according to the instructions specified on the product labels. Study products are to be dispensed by authorized site staff only to subjects enrolled in the study in accordance with the protocol.

The site must maintain adequate records documenting the receipt, use, loss, or other disposition of all the product supplies. All study products will be accounted for using the investigational/study product accountability form/record. The investigator is responsible for study product accountability, reconciliation, and record maintenance.

Subjects will return used and unused tubes of the acclimatisation toothpaste to the study site at their Baseline visit (Visit 2). Subjects will bring the used and unused tubes of their assigned study toothpaste to each of their scheduled visits to the study site, per the Schedule of Activities (<u>Table 1-1</u>); all study products will be returned at study conclusion. Study product return will be documented using the study product accountability form/record.

The accountability records must be available for inspection by the study monitor during the study. Monitoring of product accountability will be performed by the monitor during site visits and at the completion of the study.

# 6.4.1 Destruction of Study Product Supplies

At the end of the study, the investigator, or an appropriate designee, and a representative of the sponsor (study monitor) will inventory all used and unused study products and sundry items. The study product accountability record for returned study products will then be completed. All study product (used and unused) for this clinical study, will be returned for destruction to the sponsor's Clinical Supplies Department, or designated vendor, using the return instructions provided.

Detailed instructions for the return of study product/study supplies (including empty tubes) for the accountability checks and subsequent destruction will be provided by the sponsor in time for study close out visit.

Clinical Protocol

Protocol Number: 300026



# 6.5 Blinding and Allocation/Randomization

All subjects will be centrally randomized to one of the three study toothpastes using an Interactive Response Technology (IRT). Before the study is initiated, training, login information and directions for the IRT will be provided to the study site. Study products will be dispensed according to the instruction received through the IRT at the appropriate study visits.

Returned study products should not be re-dispensed to any subject.

This study is described as examiner-blind (clinical examiners will be blinded to product received). Subjects, site staff, study statistician(s), data management staff, other employees of the Sponsor (including the CRS) and vendors acting on behalf of the sponsor, who may influence study outcomes will also be blinded to product allocation. The monitors and the sponsor's Clinical Study Manager cannot be fully blinded as they will observe subjects brushing with their allocated study product while at the study site. As a matter of study conduct, including emergency unblinding events, only the investigator may learn the contents of one or more of the product codes used to allocate study product, not the clinical examiners. Given the application of IRT within this study, any such knowledge will not affect the decision to enroll a subject or influence the order in which subjects are enrolled.

To ensure the clinical examiners remain blinded throughout the study:

- Site staff involved in the dispensing of study products and supervision of on-site brushing will work in a separate area and will not be involved in any safety or product efficacy assessments.
- Clinical examiners will not be permitted in any area where study product or diaries are stored, dispensed, or in use.
- Subjects will be instructed not to remove their study product or diary from its opaque carrier bag outside of the dispensing room, while at the study site.
- Subjects will be instructed not to discuss which study product they have been assigned or usage instructions with the clinical examiners.

# 6.6 Breaking the Blind

At the initiation of the study, the study site will be instructed on the method for breaking the blind in case of emergency. The method will be an electronic process.

The electronic system will be programmed with blind-breaking instructions. In case of an emergency, the investigator has the sole responsibility for determining if unblinding of a subject's product assignment is warranted. Subject safety must always be the first consideration in making such a determination. If the investigator decides that unblinding is warranted, the investigator should make every effort to contact the sponsor prior to unblinding a subject's product assignment unless this could delay emergency treatment of the subject.

If a subject's product assignment is unblinded, the sponsor must be notified within 24 hours after breaking the blind. The date and reason that the blind was broken must be recorded in the source documentation and the eCRF, as applicable.

Any AE associated with breaking the blind must be recorded and reported as specified in this protocol. The study site may also be required be required to inform the Institutional Review Board (IRB) if the blind is broken.

Clinical Protocol

Protocol Number: 300026



# 6.7 Compliance

To facilitate compliance with product usage, subjects will be provided with a diary at Screening (Visit 1), at Baseline (Visit 2) and Week 6 (Visit 3) to record each brushing with the acclimatization toothpaste and their assigned study product, respectively.

- The diaries will provide detailed usage instructions for the subject to refer to throughout their participation in the study.
- Subjects will be instructed to note any missed/additional brushings, the reasons for any missed/additional brushings, any issues with the toothpaste used, oral problems, illnesses and any new medications/treatments in their diaries.
- Completed diaries will be reviewed by study staff at the start of each study visit. Any
  missed or additional brushings will be captured in the eCRF as protocol deviations.
  Subjects will be re-instructed in correct product usage requirements/diary completion,
  as needed.

Information recorded in the diary relating to changes in health and medications/ treatments will be reviewed by the investigator, or medically qualified designee, with the subject and transcribed into the eCRF, as appropriate (e.g., as an AE). Information related to product use should also transcribed into the eCRF, as appropriate, taking care to maintain the blind.

Subjects will be instructed to bring all tubes of toothpaste provided (used and unused) to each study visit. Study staff will perform a visual check of product usage. Any suspected over or under use will be documented in the eCRF and the subject will be re-instructed in the correct usage requirements.

To confirm subjects understood the usage instructions provided at Screening (Visit 1), they will be asked to record 2-4 brushings (one per week) during the 2-4 week acclimatisation period using their smartphone video. At Baseline (Visit 2), a designated member of the study team will check these videos to confirm compliance with the usage requirements against a checklist (Appendix 15.3). Any subjects who rinse with water during brushing with the acclimatisation toothpaste will be excluded; subjects deemed non-compliant with any other aspect of study usage requirements will be re-instructed in correct product usage.

Supervised brushings will be carried out at the study site at the end of each study visit to facilitate compliance with usage instructions. If any deviations from per protocol product usage are observed, the subject will be re-instructed of correct product usage.

Subjects will be sent reminders on WeChat to adhere to study lifestyle restrictions every 2 weeks for the duration of the study.

### 6.8 Concomitant Medications/Treatments

Any medications, treatments or vaccine (including over-the-counter or prescription medicines, vitamins, and/or herbal supplements) taken or received during the study, from signing the informed consent, must be recorded in the eCRF with indication, reason for use, unit dose, daily dose, and start and stop dates of administration. All subjects will be questioned about medications/treatments at each site visit.

Medication/treatments taken or received within 30 days of signing the informed consent form will be documented as a prior medication/treatment. Medications/treatments taken or received after signing the informed consent form will be documented as concomitant medication/treatments.

Clinical Protocol

Protocol Number: 300026



# For the Duration of the Study: Screening (Visit 1) to Subject's Last Study Visit

- Subjects should delay any non-emergency, elective dental treatments until after study completion (including dental prophylaxis).
- Should a randomized subject start a course of treatment which includes daily, regular or intermittent use of any medication, details of that medication/treatment will be recorded in the eCRF. The investigator, or their medically qualified designee, will decide if the subject can continue on the study or should be withdrawn.
- Should a subject take a medication which, in the opinion of the investigator or their medically qualified designee, could impact the subject's perception of DH (e.g., an analgesic) within 8 hours of a scheduled study visit, the medication should be recorded in the eCRF and every effort will be made to reappoint them within permitted visit tolerances (see Schedule of Activities, <u>Table 1-1</u>). The reason for re-appointment will be documented in the eCRF.

If re-appointment is not possible, the following visit specific actions should be taken:

- **Screening (Visit 1):** the subject will be withdrawn from the study. No tooth sensitivity assessments will be performed. The subject may be replaced.
- **Baseline (Visit 2):** the subject will be withdrawn from the study. No tooth sensitivity assessments will be performed. The subject will not be replaced.
- Weeks 6 & 12 (Visits 3 & 4): the subject will continue in the study. Tooth sensitivity assessments will be performed.

# 7 DISCONTINUATION OF STUDY INTERVENTION AND SUBJECT DISCONTINUATION/WITHDRAWAL

# 7.1 Subject Discontinuation/Withdrawal

A subject may withdraw from the study at any time at their own request or may be withdrawn at any time, at the discretion of the investigator or sponsor, for safety or behavioral reasons, or the inability of the subject to comply with the protocol-required schedule of study visits, procedures or lifestyle considerations.

The following circumstances require discontinuation of study product and/or premature subject withdrawal:

- Protocol violation that may impact the subject's safety
- Inability of the subject to comply with the protocol-required schedule of study visits, procedures or lifestyle considerations
- Withdrawal of informed consent
- Subject lost to follow-up
- Unblinding of the subject
- Pregnancy

If a subject is discontinued or prematurely withdraws from the study, the reason(s) for discontinuation or withdrawal and the associated date must be documented in the relevant section(s) of the eCRF.

Clinical Protocol

Protocol Number: 300026



# 7.2 Lost to Follow up

If a subject fails to return to the site for a required study visit, the site must attempt to contact the subject and reschedule the missed visit as soon as possible, counsel the subject on the importance of maintaining the assigned visit schedule and ascertain whether the subject wishes to and/or should continue in the study.

A subject will be considered lost to follow up if they repeatedly fail to return for scheduled visits and cannot be contacted by the study site. Before a subject is deemed lost to follow up, the investigator or designee must make every effort to regain contact with the subject (where possible, 3 telephone calls and, if necessary, a certified letter to the subject's last known mailing address or local equivalent methods). All contact attempts should be documented in the eCRF. If contact is made, the investigator or designee should inquire about the reason for withdrawal, request that the subject return all study products provided and, if appropriate, request the subject return for a final visit and follow-up with the subject regarding any unresolved AEs.

Final safety assessments may be carried out when the subject returns to the study site, at the investigator's discretion, which may include an oral examination.

Should the subject be unreachable, they will be considered to have withdrawn from the study and lost to follow up.

Lack of completion of all or any of the early termination procedures will not be viewed as protocol deviations provided the subject's safety was preserved.

If the subject withdraws from the study and withdraws consent for disclosure of future information, no further evaluations should be performed and no additional data should be collected. The sponsor may retain and continue to use any data collected before such withdrawal of consent.

### 8 STUDY PROCEDURES

This section lists the procedures to be completed at each planned study visit. The timing of each procedure is listed in the Schedule of Activities section (<u>Table 1-1</u>).

Adherence to the study design requirements, including all procedures are essential and required for study conduct.

# 8.1 Visit 1/Screening

The following procedures and assessments will be completed by the investigator, or a suitably qualified/experienced designee, and the clinical examiners, 14-28 days prior to randomisation to study product. Where practically feasible, they should be completed in the order listed below. Data collected will be recorded in the eCRF.

### 8.1.1 Informed Consent

The investigator, or designee, must obtain informed consent from each subject participating in the study after adequate explanation of the aims, methods, objectives, and potential hazards of the study. Study information will be communicated to the subjects by the investigator, or designee, and by interactive video which will also be sent to the subjects via WeChat for their own reference. After signing the ICF, subjects will be asked to complete a knowledge check (a quiz) to ensure key information and study expectations are understood. If the subject answers one or more questions incorrectly, the study information will be re-explained and the subject
Clinical Protocol

Protocol Number: 300026



will be asked to complete knowledge check again. If subjects are not able to understand the study information, they will be excluded.

A list of ingredients in the toothpastes to be used during the study will be provided to each subject during the consent process to enable them to confirm they are not aware of any allergy or hypersensitivity to any of the ingredients listed.

The investigator, or designee, must explain to the subjects that they are completely free to refuse to enter the study or to withdraw from it at any time.

Appropriate forms for documenting consent will be provided by either the investigator or the sponsor. Two copies of the ICF will be signed and dated by the subject; the subject will retain one copy, the other will be kept at site. The time the ICF was signed by the subject will be recorded on the ICF; AEs will be captured from that time. The investigator, or designee, will sign and date each copy of the ICF after the subject has signed to confirm that the consent process was completed correctly. The date and time subject received the ICF and signed the ICF will be recorded in the eCRF.

If new information becomes available during the course of the study that could affect willingness to participate, each participating subject will receive a copy of the new information and be re-consented into the study (2 copies as before). Each subject will be provided with a copy of the signed and dated amended consent form. The date and time of re-consent will be recorded in the eCRF.

After signing the ICF, subjects will undergo the screening assessments to confirm they meet the subject selection criteria for the study. If the subject is confirmed eligible by the investigator or designee to participate, the subject will be considered enrolled in the study.

#### 8.1.2 Demographics

The following demographic information will be recorded in the CRF: year of birth, sex (male or female) and race.

#### 8.1.3 Check of the WeChat Application

Subjects will be also asked to show study staff their mobile phone to confirm the WeChat application is installed. Subjects who do not have WeChat and are not willing to install it while at the study site will be excluded.

#### 8.1.4 DH Screening Questionnaire

Subjects will complete a screening questionnaire (<u>Appendix 15-2</u>) to confirm self-reported DH symptoms. Subjects who report experiencing DH symptoms only 'several times a month', 'once a month' or 'less than once a month' will be excluded from the study.

#### 8.1.5 Review of Oral Care Products

Subjects will be required to bring their current oral care products to the Screening visit for study staff to confirm the <u>absence of known anti-sensitivity ingredients</u> and DH relief claims on the packaging. Presence/absence of fluoride will also be documented in the eCRF.

Subjects who are currently using anti-sensitivity oral care product(s) will be excluded.

Subjects will also be asked about the oral care products they have been using in the last 8 weeks; those who report using anti-sensitivity product(s) in the previous 8 weeks will also be excluded.

Clinical Protocol

Protocol Number: 300026



#### 8.1.6 Review of Brushing Habits

Subjects will be asked to describe their typical oral care routine. Subjects who habitually rinse with water during toothbrushing will be excluded.

# 8.1.7 Medical History and Prior Medication/Treatment

The following will be documented in the eCRF:

- Details of relevant medical history and recent surgery (within the last year), including allergies and drug sensitivities.
- Pregnancy status (self-reported by female subjects only).
- Prior medications/treatments, including prescription and non-prescription drugs, dietary supplements and herbal remedies, taken in the last 30 days.

#### 8.1.8 Clinical Examinations and Assessments

Prior to commencing the clinical examinations and assessments, subjects will be shown how to complete a VAS (Section 9.1.3).

The following clinical examinations will be completed as described in <u>Study Assessments</u> and the findings recorded in the eCRF. To facilitate subject flow, source documents can be used to record the eligible teeth and DH assessments for later transcription into the eCRF (transcription from source documents must be completed within 5 days of recording the data for each subject).

- OST examination
- OHT examination
- Clinical assessment of incisors, canines and pre-molars for dentition exclusions, EAR, MGI (adjacent to the test area only) and clinical mobility to identify eligible teeth for DH assessment (as described in Section 9.1).
- Clinical assessment of tactile sensitivity (tactile threshold (g)) for each eligible tooth (no dentition exclusions, presence of EAR, MGI = 0 adjacent to the test area only, clinical mobility = 0).
- Clinical assessment of evaporative (air) sensitivity (Schiff sensitivity score [examiner assessed], followed by VAS [subject completed]) for each eligible tooth with a tactile threshold of ≤ 20g.

There should be at least a 5-minute break between completing the tactile assessments and starting the evaporative (air) assessments.

To prepare for the Baseline visit, the clinical examiners will confirm those teeth which are eligible for ongoing DH assessment at Baseline (Visit 2).

• 'Eligible teeth identified at Screening' (<u>Table 4-1</u>): incisors, canines and pre-molars with none of the study-specific dentition exclusions, which meet EAR, MGI adjacent to the test area <u>only</u> and mobility inclusion criteria, and record a qualifying tactile threshold of  $\leq 20$  g and a qualifying Schiff sensitivity score of  $\geq 2$  at Screening (Visit 1).

#### 8.1.9 Inclusion/Exclusion Criteria

Information relating to all inclusion and exclusion criteria will be completed in the eCRF.

Clinical Protocol

Protocol Number: 300026



#### 8.1.10 Subject Eligibility

The investigator, or medically qualified designee, will review the inclusion/exclusion criteria to confirm subject eligibility to participate in the study; this will be documented in the eCRF.

Note: In addition to meeting all other study requirements, only those subjects with a minimum of two eligible teeth with a qualifying tactile threshold  $\leq 20$  g and a qualifying Schiff sensitivity score  $\geq 2$  can continue on the study.

To prepare for study participation, enrolled subjects will be instructed in the <u>Lifestyle Guidelines</u> and <u>Concomitant Medications/Treatments</u> requirements of the study (as already detailed in the ICF and described during the consent process). Adherence to the requirements of the study protocol is essential for successful study conduct.

#### 8.1.11 Supervised Brushing with Acclimatization Toothpaste

Enrolled subjects will be provided with the acclimatization toothpaste, a toothbrush, a timer, rinsing cups and a diary to use during the acclimatization period.

Staff will describe the toothpaste usage instructions to the subject and demonstrate covering the full brush head with a ribbon of toothpaste. Staff will then supervise the subject carrying out first their first brushing with the acclimatization toothpaste and recording the first use in their diary.

Any deviation from the product usage instructions will be captured as a protocol deviation in the eCRF and the subject will be reminded of the correct directions for use. Dispensing of the acclimatization toothpaste and completion of the supervised first brushing will also be documented in the eCRF.

Spontaneously reported AEs, and any AEs elicited by asking subjects to respond to a non-leading question, such as 'How do you feel?', on completion of the supervised brushing with the acclimatization toothpaste will be recorded in the eCRF.

Staff will remind subjects to bring their acclimatisation products to their next study visit and to note any changes in health, medications or treatments in their diary (or report such changes to study staff between visits using the contact numbers provided or inform the staff at their next visit, if preferred).

#### 8.2 Study Period

#### 8.2.1 Visit 2 (Baseline/Day 1)

The following procedures and assessments will be completed by the investigator, or a suitably qualified/experienced designee and the clinical examiners. Where practically feasible, they should be completed in the order listed below. All data collected should be recorded in the eCRF.

#### 8.2.1.1 Compliance Checks

Complete visual checks of returned acclimatization toothpaste, review completed diary and watch the brushing videos (using the Video Compliance Checklist (<u>Appendix 15.3</u>) to help determine compliance). Subjects seen to rinse with water while brushing with the acclimatization toothpaste during review of their brushing compliance videos will be excluded.

Clinical Protocol

Protocol Number: 300026



Record any suspected over or under use and the number of any missed or additional brushings in the eCRF. Any deviation from the product usage instructions or missed brushing videos will be captured as protocol deviations in the eCRF and subjects will be re-instructed in the correct directions for use.

Do not return the acclimatization toothpaste, toothbrush or completed diary to the subject.

#### 8.2.1.2 Changes in Medical History and Concomitant Medications/Treatments

Staff will ask subjects if there have been any changes in their health, concomitant medications and non-drug treatments/procedures. All changes will be documented in the eCRF.

Spontaneous reporting of AEs and those elicited by asking subjects to respond to a non-leading question, such as 'How do you feel?', will be assessed and any AEs recorded in the eCRF.

Any AEs and/or changes in medications/treatments identified during review of the completed diary will also be recorded in the eCRF.

#### 8.2.1.3 Subject Adherence and Continuance

Confirm subject adherence to the requirements of the protocol and document their continuance in the eCRF. Record any deviations from study requirements in the eCRF.

#### 8.2.1.4 Clinical Examinations and Assessments

Prior to commencing the clinical examinations and assessments, subjects will be reminded how to complete a VAS (Section 9.1.3).

The following clinical examinations will be completed as described in <u>Study Assessments</u> and the findings recorded in the eCRF. To facilitate subject flow, source documents can be used to record the DH assessments for later transcription into the eCRF (transcription from source documents must be completed within 5 days of recording the data for each subject).

- OST examination
- Clinical assessment of tactile sensitivity (tactile threshold (g)) for each *eligible tooth identified at Screening* (eligibility criteria described in Section 8.1.8 and Table 4-1).
- Clinical assessment of evaporative (air) sensitivity (Schiff sensitivity score [examiner assessed], followed by VAS [subject completed]) for each eligible tooth identified at Screening with a <u>Baseline</u> tactile threshold of ≤ 20g.

There should be at least a 5-minute break between completing the tactile assessments and starting the evaporative (air) assessments.

Subjects must have at least two eligible teeth with the qualifying tactile threshold  $\leq 20$  g and qualifying Schiff sensitivity score  $\geq 2$  at both Screening <u>and</u> Baseline, and VAS  $\geq 40$  mm at Baseline to continue.

#### 8.2.1.5 Selection of Test Teeth

The procedure for selecting test teeth is summarised in <u>Table 4-1</u>

The clinical examiner responsible for 'Schiff' assessments will examine all qualifying teeth both at Screening and Baseline to identify two 'test teeth' for DH assessment at subsequent study visits. The identity of the two test teeth will be recorded in the eCRF. Subjects with fewer than two suitable test teeth will be discontinued.

Property of GSK Consumer Healthcare - Confidential

Clinical Protocol

Protocol Number: 300026



- Test teeth can only be selected from eligible teeth with the 'qualifying' levels of DH:
  - Tactile threshold  $\leq 20$  g at Screening (Visit 1) and Baseline (Visit 2).
  - Schiff sensitivity score  $\geq 2$  at Screening (Visit 1) and Baseline (Visit 2).
  - VAS  $\geq$  40 mm at Baseline (Visit 2).
- Each test tooth must have the <u>same</u> Schiff sensitivity score at Screening <u>and</u> Baseline.

| <b>Screening</b> Schiff sensitivity score = 2 <u>and</u> <b>Baseline</b> Schiff sensitivity score = 2 |
|---|
| OR |
| <b>Screening</b> Schiff sensitivity score = 3 <u>and</u> <b>Baseline</b> Schiff sensitivity score = 3 |

# 8.2.1.6 Subject Eligibility

The investigator, or medically qualified designee, will review the inclusion/exclusion criteria and verify the presence of two test teeth which meet all study criteria before confirming each subject's suitability to continue in the study; eligibility will be documented in the eCRF.

#### 8.2.1.7 Stratification and Randomization

Eligible subjects will be stratified to one of two strata as described in <u>Section 5.4</u>. Subject stratum will be entered directly into the eCRF. Each subject will be assigned a randomisation number from their designated stratum in ascending numerical order, and as each subject is determined to be fully eligible. The randomized toothpaste code will be entered directly into the eCRF.

#### 8.2.1.8 Supervised Brushing with Study Toothpaste

Randomised subjects will be provided with their allocated study toothpaste, a new toothbrush, more rinsing cups and a new diary.

Toothpaste usage instructions will be re-described, and those subjects randomized to the test toothpaste will be shown the location of their two 'test teeth' within the mouth (using a tooth diagram/model and a mirror, as appropriate). Staff will then supervise the subject carrying out first the first brushing with their study toothpaste and recording the first use in their diary. A brushing video will be also shared with the subjects via WeChat according to their allocated study toothpaste.

Any deviation from the product usage instructions will be captured as a protocol deviation in the eCRF and the subject will be reminded of the correct directions for use. Dispensing of study toothpaste and completion of the supervised first brushing will also be documented in the eCRF.

Spontaneously reported AEs, and any AEs elicited by asking subjects to respond to a non-leading question, such as 'How do you feel?', on completion of the supervised brushing with the study toothpaste will be recorded in the eCRF.

Randomized subjects will be re-instructed of the <u>Lifestyle Guidelines</u> and <u>Concomitant Medications/Treatments</u> requirements of the study. Staff will remind them to bring their study products to their next study visit and to note any changes in health, medications or treatments in their diary (or report such changes to study staff between visits using the contact numbers provided or inform the staff at their next visit, if preferred).

Clinical Protocol

Protocol Number: 300026



#### 8.2.2 Visit 3 (Week 6/Day 43 $\pm$ 4) and Visit 4 (Week 12/Day 85 $\pm$ 4)

The following procedures and assessments will be completed by the investigator, or a suitably qualified/experienced designee and the clinical examiners. Where practically feasible, they should be completed in the order listed below. All data collected should be recorded in the eCRF.

#### 8.2.2.1 Compliance Checks

Complete visual checks of returned study toothpaste and review completed diary. Record any suspected over or under use and the number of any missed or additional brushings in the eCRF.

Any deviation from the product usage instructions will be captured as protocol deviations in the eCRF and subjects will be re-instructed in the correct directions for use.

Week 6 (Visit 3): Return the study toothpaste to the subject; retain the used toothbrush and completed 'Week 6' diary at site. Dispense new diary card and new toothbrush.

Week 12 (Visit 4): Retain the study toothpaste, toothbrush and completed 'Week 12' diary.

### 8.2.2.2 Changes in Medical History and Concomitant Medications/Treatments

Staff will ask subjects if there have been any changes in their health, concomitant medications and non-drug treatments/procedures. All changes will be documented in the eCRF.

Spontaneous reporting of AEs and those elicited by asking subjects to respond to a non-leading question, such as 'How do you feel?', will be assessed and any AEs recorded in the eCRF.

Any AEs and/or changes in medications/treatments identified during review of the completed diary will also be recorded in the eCRF.

#### 8.2.2.3 Subject Adherence and Continuance

Confirm subject adherence to the requirements of the protocol and document their continuance in the eCRF. Record any deviations from study requirements in the eCRF.

#### 8.2.2.4 Clinical Examinations and Assessments

Prior to commencing the clinical examinations and assessments, subjects will be reminded how to complete a VAS (Section 9.1.3).

The following clinical examinations will be completed as described in <u>Study Assessments</u> and the findings recorded in the eCRF. To facilitate subject flow, source documents can be used to record the DH assessments for later transcription into the eCRF (transcription from source documents must be completed within 5 days of recording the data for each subject).

- OST examination
- Week 12 (Visit 4) only: OHT examination
- Clinical assessment of tactile sensitivity (tactile threshold (g)) for the two test teeth only.
- Clinical assessment of evaporative (air) sensitivity (Schiff sensitivity score, followed by VAS) for the two test teeth only.

There should be at least a 5-minute break between completing the tactile assessments and starting the evaporative (air) assessments.

Clinical Protocol

Protocol Number: 300026



### 8.2.2.5 Supervised Brushing with Study Toothpaste

#### Week 6 (Visit 3) only:

Subjects will be provided with a new toothbrush and a new diary; staff will supervise each subject completing another on-site brushing with their study toothpaste and recording this use in their diary.

Any deviation from the product usage instructions will be captured as a protocol deviation in the eCRF and the subject will be reminded of the correct directions for use. Completion of the 'Week 6' supervised brushing will also be documented in the eCRF.

Spontaneously reported AEs, and any AEs elicited by asking subjects to respond to a non-leading question, such as 'How do you feel?', on completion of the supervised brushing with the study toothpaste will be recorded in the eCRF.

Subjects will be re-instructed of the <u>Lifestyle Guidelines</u> and <u>Concomitant Medications/</u>
<u>Treatments</u> requirements of the study. Staff will remind them to bring their study products to their next study visit and to note any changes in health, medications or treatments in their diary (or report such changes to study staff between visits using the contact numbers provided or inform the staff at their next visit, if preferred).

#### Week 12 (Visit 4) only:

No supervised brushing.

### 8.3 Study Conclusion

The Study Conclusion page of the eCRF will be completed for all subjects whether or not they complete all study procedures (e.g., if they are discontinued from the study early). If the subject is discontinued early, at any point during the study, the primary reason for withdrawal should be recorded on the Study Conclusion page.

For subjects who attend all study visits, the Study Conclusion page of the eCRF will be completed at Visit 4. Staff will remind each subject to inform the site if they experience any change in health, medications or treatments in the next 5 days (i.e., in the 5 days following their last use of study product).

If a subject has any clinically significant, study-related abnormalities or AEs at the end of the study, the sponsor's medical monitor (or designated representative) should be notified and, the subject may be asked to return for a follow-up visit to ensure any issue is resolved or deemed not clinically significant.

#### 8.4 Follow-up Visit / Phone Call

The study site may contact a subject to follow up an AE post-study completion/withdrawal and, in some circumstances, request they return to the site for additional follow-up visits (final safety assessments). At the discretion of the investigator, or medically qualified designee, additional oral examinations may be carried out at such visits.

#### 9 STUDY ASSESSMENTS

Every effort should be made to ensure the protocol-required examinations and assessments are completed as described. However, it is anticipated that from time to time there may be circumstances, outside of the investigator's control, that may make it unfeasible to complete an



examination or assessment. In these cases, the investigator must take all steps necessary to ensure the safety and well-being of the subject. When a protocol-required examination or assessment cannot be performed, the investigator (or designee) will document the reason for the missed procedure as a protocol deviation and any corrective and preventative actions they have taken to ensure that required processes are adhered to as soon as possible. The Sponsor must be informed of any missed examinations or assessments in a timely manner.

# 9.1 Screening Assessments

Screening assessments will be performed by appropriately trained staff/clinical examiners (dentists) at the times, and in the order, defined in the Study Procedures section of this protocol.

The eligibility of each tooth will be assessed against the inclusion/exclusion criteria and recorded in the eCRF.

#### 9.1.1.1 Erosion, Abrasion and Recession (EAR)

The facial surfaces of all incisor, canine and pre-molar teeth (<u>Figure 9-1</u>) that do not present any of the general dentition exclusion criteria, or specific dentition exclusion criteria for eligible teeth, will be examined for signs of cervical EAR (Addy, 2000).



Figure 9-1 Dental Nomenclature. (Dempsey and Townsend, 2001)

#### 9.1.1.2 Modified Gingival Index (MGI)

The MGI is a non-invasive visual assessment of gingival health (<u>Lobene</u>, <u>1986</u>). MGI will be assessed for incisor, canine and pre-molar teeth exhibiting none of the dentition exclusions and facial/cervical EAR. MGI should be scored for the facial gingiva, <u>directly adjacent to the area of exposed dentine</u> (i.e., the test area) <u>only</u>.

Eligible teeth will have a MGI of zero (0) directly adjacent to the test area.

| Score | Description |
|---|---|
| 0 | Absence of inflammation |
| 1 | Mild inflammation; slight change in colour, little change in colour; little change in texture of any portion of the marginal or papillary gingival unit. |
| 2 | Mild inflammation; criteria as above but involving the entire marginal or papillar gingival unit. |
| 3 | Moderate inflammation; glazing, redness, oedema, and/or hypertrophy of the marginal or papillary gingival unit. |
| 4 | Severe inflammation; marked redness, oedema and/or hypertrophy of the marginal or papillary gingival unit, spontaneous bleeding, congestion, or ulceration. |

Clinical Protocol

Protocol Number: 300026



#### 9.1.1.3 Clinical Mobility

Clinical mobility will be assessed for incisor, canine and pre-molar teeth exhibiting none of the dentition exclusions, with facial/cervical EAR and a MGI = 0 adjacent to the test area only, using a modification of the Miller Index (<u>Laster</u>, 1975).

#### Eligible teeth will have clinical mobility = 0.

| Degree | Description |
|---|---|
| 0 | No movement or mobility of the crown of the tooth < 0.2mm in a horizontal direction |
| 1 | Mobility of the crown of the tooth 0.2 - 1mm in a horizontal direction |
| 2 | Mobility of the crown of the tooth exceeding 1mm in a horizontal direction |
| 3 | Mobility of the crown of the tooth in a vertical direction as well. |

#### 9.1.2 Qualifying Tactile Sensitivity

The tactile sensitivity of incisor, canine and pre-molar teeth (<u>Figure 9-1</u>) exhibiting none of the dentition exclusions, and meeting the EAR, MGI (adjacent to the test area only) and clinical mobility criteria, will be assessed using a constant pressure probe (Yeaple probe (<u>Polson et al.</u>, <u>1980</u>). The probe tip will be placed perpendicular to the facial surface of the tooth and drawn slowly across the exposed dentine to ensure application of the stimulus across the potentially 'sensitive' area.

After each application of the tactile stimulus, the subject will be asked to indicate whether they experienced any pain or discomfort. The examiner will tell the subject to only respond 'yes' if they feel PAIN or DISCOMFORT when the probe is applied to their tooth. 'Yes' and 'no' are the only acceptable answers. The subject may respond 'yes' if they feel pressure. The examiner will remind them, as needed, that they will feel pressure each time the probe is in contact with the tooth but they should only respond 'yes' if they feel pain or discomfort. The gram setting which elicits the two consecutive 'yes' responses will be recorded as the tactile threshold (g) in the source document. At Screening, the upper force setting will be 20g.

- For a tooth to qualify at Screening, it must have a tactile threshold  $\leq 20g$ .
- If no sensitivity is found at the upper force setting, the tactile threshold will be recorded as > 20g and the tooth will be disqualified from further testing.

If a subject fails to give a definite answer, the examiner will re-prompt them to provide a 'yes' or 'no' response. If their uncertainty continues, this should be recorded on the source document. and the next stimulus should be at the next step in the upward direction. If the subject continues to be unsure, or the examiner is unsure of the reliability of their response, the examiner may opt to re-probe at the same force setting (indicated to the scribe by a non-verbal signal, e.g., a hand gesture) or move to the next force setting (10g increase). If the examiner considers the subject's 'yes' response may be between gram settings, a conservative approach should always be adopted, and the lower (more 'severe') tactile threshold (g) recorded.

The examiner will generally make the force setting adjustments (this can also be done by an assistant/scribe); the scribe will record the micro-amperage setting and subject's responses in the source document.

#### Calibration of the Yeaple Probe:

The Yeaple probe will be calibrated by an appropriately trained member of the study staff (typically the clinical examiner or their assistant/scribe) before use on each day subjects are

Property of GSK Consumer Healthcare - Confidential

Clinical Protocol

Protocol Number: 300026



assessed. The microamp settings may vary from day to day (partly due to battery power consumption), but the difference should not be significant. Thus, previous probe settings can serve as a guide. Calibration should start at the lowest microamp setting and then increase. Either calibration method described below is acceptable.

- Method 1 ('Water Cup'): The Yeaple probe is fixed to a clamp attached to a ring stand so that the probe tip is vertical. A small paper cup attached with cotton thread is balanced over the end of the Yeaple probe, without the probe tripping. The probe dial is set to the microamp setting and water is fed into the paper cup using a dropper until the probe trips. The gram setting is recorded and the Yeaple probe reset to the next microamp value. The procedure is repeated until data has been collected to more than 80 g.
- **Method 2:** The Yeaple probe is fixed to a clamp attached to a ring stand so that the top is perpendicular to the pan of an ohaus dial-o-gram<sup>®</sup> balance or equivalent. The probe tip is positioned to just touch the pan when the balance is set at zero grams. The probe dial is set to the microamp setting and the gram setting is increased on the balance until the probe trips. The gram setting is recorded and the Yeaple probe reset to the next microamp value.

The data are plotted, and the points connected with line segments in order to interpolate the micro-amp values equivalent to 10, 20, 30, 40, 50, 60, 70 and 80 g. This calibration should be repeated three times, and the average of the three used for the day's settings. The settings will be recorded on the Yeaple probe calibration record (along the probe's serial number) which will serve as the force setting guide for that day's examinations.

# 9.1.3 Qualifying Evaporative (Air) Sensitivity

Evaporative (air) sensitivity will be assessed on the facial surfaces of incisor, canine and premolar teeth (Figure 9-1) which exhibit none of the dentition exclusions, and meet the EAR, MGI (adjacent to the test area only), clinical mobility and tactile threshold ( $\leq$  20g) criteria. Assessment will start a minimum of 5 minutes after the tactile assessments have completed. The assessment will be made by directing a 1-second application of air from a standard dental syringe held perpendicular to the tooth surface, approximately 1-2 mm coronal to the gingival margin, and from a distance of approximately 1 cm. The dental examiner will take appropriate measures to isolate the tooth surface to prevent stimulation of adjacent teeth or surrounding soft tissue.

Subject response to the stimulus will be evaluated using the Schiff sensitivity scale (Schiff, 1994). This is an examiner-based index, scored immediately following administration of the evaporative (air) stimulus. The scale focuses on a combination of specific, observable, physical, behavioural and verbal responses from the subject, which may facilitate discrimination.

| Score | Description |
|---|---|
| 0 | Subject does not respond to air stimulation |
| 1 | Subject responds to air stimulus but does not request discontinuation of stimulus |
| 2 | Subject responds to air stimulus and requests discontinuation or moves from stimulus |
| 3 | Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus |

Clinical Protocol

Protocol Number: 300026



If the clinical examiner assesses the subject response to be between scores, a conservative approach should always be adopted, and the higher (more 'severe') score recorded.

After the clinical examiner has communicated each Schiff sensitivity score to the scribe (nonverbally), the subject will rate the intensity of their response to the evaporative (air) stimulus using a 100 mm VAS (example below). The clinical examiner and the subject should be blinded to their respective scores.



A trained member of staff will measure the distance (mm) from zero (0) to the left of the line marked by the subject and record this value in the eCRF.

- For a tooth to qualify at Screening, it must have a tactile threshold  $\leq 20g$  and a Schiff sensitivity score  $\geq 2$ .
- If Schiff sensitivity score = 0 or 1, the tooth will be disqualified from further testing (the subject's VAS response will still be recorded).

# 9.2 Dentine Hypersensitivity Efficacy Assessments

The following product efficacy assessments will be performed by appropriately trained clinical examiners (who are blind to product received), at the times and in the order defined in the <u>Study Procedures</u> section of this protocol.

The same examiner will be responsible for a given DH assessment (tactile or evaporative (air) sensitivity) throughout the study (Visit 1 to Visit 4).

#### 9.2.1 Tactile Sensitivity Assessment (Yeaple Probe)

#### **Baseline (Visit 2):**

The tactile sensitivity of all *eligible teeth identified at Screening* (Visit 1) will be assessed for all enrolled subjects. The tactile stimulus will be administered, and subject response recorded as described in Section 9.1.2. At Baseline, the upper force setting will be 20g.

- For a tooth to 'qualify' at Baseline, it must have a tactile threshold  $\leq 20g$ .
- If no sensitivity is found at the upper force setting, the tactile threshold will be recorded as > 20g and the tooth will be disqualified from further testing.

**Note:** 'Eligible teeth identified at Screening' are defined as incisors, canines and pre-molars with none of the study-specific dentition exclusions, which meet the EAR, MGI (adjacent to the test area only) and mobility inclusion criteria, and record a qualifying tactile threshold of  $\leq$  20g and a qualifying Schiff sensitivity score of  $\geq$  2 at Screening (Visit 1).

#### Week 6 (Visit 3) & Week 12 (Visit 4):

The tactile sensitivity of the two test teeth identified by the clinical examiners at Baseline (Visit 2) will be assessed for all randomized subjects. The tactile stimulus will be administered, and subject response recorded as described in Section 9.1.2.

Clinical Protocol

Protocol Number: 300026



At Week 6 and Week 12, the upper force setting will be 80g. The gram setting, which elicits two consecutive 'yes' responses, will be recorded as the tactile threshold (g). If no sensitivity is found, the tactile threshold should be recorded as >80g.

#### 9.2.2 Evaporative (Air) Sensitivity Assessments

#### **Baseline (Visit 2):**

The evaporative (air) sensitivity of all *eligible teeth identified at Screening* (Visit 1), with a Baseline tactile threshold  $\leq 20$ g, will be assessed for all enrolled subjects. The evaporative (air) stimulus will be administered, and subject response (Schiff sensitivity score, followed by VAS) recorded as described in Section 9.1.3. Assessment will start a minimum of 5 minutes after the tactile assessments have completed.

- For a tooth to 'qualify' at Baseline, it must have a tactile threshold  $\leq 20g$ , a Schiff sensitivity score of  $\geq 2$  and a VAS  $\geq 40$  mm.
- If Schiff sensitivity score is < 2, the tooth will be disqualified from further testing.

#### Week 6 (Visit 3) & Week 12 (Visit 4):

The evaporative (air) sensitivity of the <u>two test teeth</u> identified by the clinical examiners at Baseline (Visit 2) will be assessed for all randomized subjects. The evaporative (air) stimulus will be administered, and subject response (Schiff sensitivity score, followed by VAS) recorded as described in Section 9.1.3.

### 9.3 Safety and Other Assessments

The following safety assessments will be performed by appropriately trained clinical examiners, at the times and in the order defined in the Study Procedures section of this protocol.

#### 9.3.1 Oral Soft Tissue (OST) Examination

The OST examination will be accomplished by direct observation and palpation, using retraction aids as appropriate, and will include examination of the labial mucosa (including lips), buccal mucosa, mucogingival folds, gingival mucosa, hard palate, soft palate, tonsillar area, pharyngeal area, tongue, sublingual area, submandibular area and salivary glands. The results of the examination will be recorded in the eCRF as either 'normal' or 'abnormal'; details of any abnormalities will be documented in the eCRF.

Any observation that changes from 'normal' to 'abnormal', or worsens, from the OST examination completed at Screening will be recorded as an AE.

#### 9.3.2 Oral Hard Tissue (OHT) Examination

The OHT examination will be accomplished by direct observation, using retraction aids as appropriate, and will identify enamel irregularities, tooth fractures, grossly carious lesions/gross decay, defective/faulty restorations (all direct & indirect restorations including fixed/removal prostheses), non-carious tooth surface loss (abrasion, attrition, abfraction and erosion), any other hard tissue irregularities (e.g., hypo/hypermineralisation, decalcification) and significant tooth staining. Observations will be listed as 'absent' or 'present'; conditions noted as 'present' will be described in the eCRF. Any observation that changes from 'absent' to 'present', or worsens, from the OHT examination completed at Screening will be recorded as an AE.

Clinical Protocol

Protocol Number: 300026



The presence of any implants, fixed or removable dentures, fixed or removable orthodontic braces/bands, fixed orthodontic retainers, full crowns or veneers will be recorded, along with evidence of gross intra-oral neglect or the need for extensive dental therapy.

The OHT examination is also used to assess the dentition against the general and specific dentition exclusions described in Section 5.3 (Exclusion Criteria 25, 26, 27, 28 and 29 a) to f)).

#### 9.3.3 Pregnancy

This clinical study will evaluate toothpastes classified as general goods in China. Sponsor studies in which no drug is utilized do not require pregnancy testing.

Female subjects will provide verbal confirmation of pregnancy status at Screening (Visit 1) and will be asked to inform study staff immediately should this change at any point during the study.

Female subjects who are pregnant or intending to become pregnant during the study (self-reported) will be excluded.

#### 10 ADVERSE EVENT AND SERIOUS ADVERSE EVENTS

The investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study product or the study, or that caused the subject to discontinue the study product or study.

# 10.1 Definition of an Adverse Event (AE)

An AE is any untoward medical occurrence in a clinical study subject, temporally associated with the use of a study product including any washout or lead-in product (or medical device), whether or not considered related to the study product, including any washout or lead-in product (or medical device).

NOTE: An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study product including any washout or lead-in product (or medical device).

#### **Events Meeting the AE Definition:**

- Any abnormal laboratory test results (hematology, clinical chemistry, or urinalysis) or
  other safety assessments (e.g., electrocardiogram (ECG), radiological scans, vital sign
  measurements), including those that worsen from baseline, considered clinically
  significant in the medical and scientific judgment of the investigator (i.e., not related to
  progression of underlying disease).
- Exacerbation of a chronic or intermittent pre-existing condition including either an increase in frequency and/or intensity of the condition.
- New conditions detected or diagnosed after study product administration even though it may have been present before the start of the study.
- Signs, symptoms, or the clinical sequelae of a suspected drug-drug interaction.
- Signs, symptoms, or the clinical sequelae of a suspected overdose of either study product or a concomitant medication. Overdose per se will not be reported as an AE/SAE unless it is an intentional overdose taken with possible suicidal/self-harming intent. Such overdoses should be reported regardless of sequelae.

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH



Protocol Number: 300026



• 'Lack of efficacy' or 'failure of expected pharmacological action' per se will not be reported as an AE. Such instances will be captured in the efficacy assessments. However, the signs, symptoms, and/or clinical sequelae resulting from lack of efficacy will be reported as AE if they fulfill the definition of an AE.

# **Events NOT meeting the AE definition:**

- Any clinically significant abnormal laboratory findings (if applicable) or other abnormal safety assessments which are associated with the underlying disease, unless judged by the investigator to be more severe than expected for the subject's condition.
- The disease/disorder being studied or expected progression, signs, or symptoms of the disease/disorder being studied, unless more severe than expected for the subject's condition.
- Medical or surgical procedure (e.g., endoscopy, appendectomy) is not the AE. The condition that leads to the procedure is an AE (e.g., appendicitis).
- Situations where an untoward medical occurrence did not occur (social and/or convenience admission to a hospital).
- Anticipated day-to-day fluctuations of pre-existing disease(s) or condition(s) present or detected at the start of the study that do not worsen.

# 10.2 Definition of a Serious Adverse Event (SAE)

A serious adverse event (SAE) is a particular category of an AE where the adverse outcome is serious. If an event is not an AE per definition above, then it cannot be an SAE, even if serious conditions are met (e.g. hospitalization for signs/symptoms of the disease under study, death due to progression of disease).

A serious adverse event is any untoward medical occurrence at any dose that:

#### • Results in death

#### • Is life-threatening

- The term 'life-threatening' in the definition of 'serious' refers to an event in which the subject was at risk of death at the time of the event. It does not refer to an event, which hypothetically might have caused death, if it were more severe.

#### • Requires inpatient hospitalization or prolongation of existing hospitalization

- In general, hospitalization signifies that the subject has been detained (usually involving at least an overnight stay) at the hospital or emergency ward for observation and/or treatment that would not have been appropriate in the physician's office or outpatient setting. Complications that occur during hospitalization are AEs. If a complication prolongs hospitalization or fulfills any other serious criteria, the event is serious. When in doubt as to whether 'hospitalization' occurred, or was necessary, the AE should be considered serious.
- Hospitalization for elective treatment of a pre-existing condition that did not worsen from baseline is not considered an AE.

#### • Results in persistent or significant disability/incapacity

- The term disability means a substantial disruption of a person's ability to conduct normal life functions.

Protocol Number: 300026



- This definition is not intended to include experiences of relatively minor medical significance such as uncomplicated headache, nausea, vomiting, diarrhea, influenza, and accidental trauma (e.g., sprained ankle) which may interfere with or prevent everyday life functions but do not constitute a substantial disruption

#### • Results in congenital anomaly/birth defect

#### • Other situations:

- Medical or scientific judgment should be exercised in deciding whether SAE reporting is appropriate in other situations such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition. These events should usually be considered serious.
- Examples of such events include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, or development of drug dependency or drug abuse.

**Note:** Classification of an AE as 'serious' is based on the outcome of the event and is a factor in determining reporting requirements.

# 10.3 Time Period and Frequency for Collecting AE and SAE Information

All AEs, and therefore all SAEs, will be collected immediately after a subject provides consent to participate in the study by the completion (signature) of the ICF and until 5 days following last administration of the study product (or last study procedure).

Medical occurrences that began before obtaining informed consent will be recorded in the Medical History/Current Medical Conditions section of the eCRF, not the AE section.

Details recorded by the subject on a diary or similar document that meet the definition of an AE must also be discussed with the subjects and transcribed in the AE section of the eCRF.

All SAEs will be recorded and reported to the sponsor or designee immediately and under no circumstance should this exceed 24 hours. The investigator will submit any updated SAE data to the sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek AEs or SAEs after the conclusion of the study participation. However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and they consider the event to be reasonably related to the study product or study participation, the investigator must promptly notify the sponsor.

# 10.4 Reporting Procedures

The investigator and any designees are responsible for detecting, documenting and reporting events that meet the definition of an AE and remain responsible for following up on AEs that are serious, considered related to the study product(s), participation in the study, or a study procedure, or that caused the subject to discontinue the study product or study.

Clinical Protocol

Protocol Number: 300026



Spontaneous reporting of AEs and those elicited by asking subjects to respond to non-leading question, such as 'How do you feel?', will be assessed and any AEs recorded in the eCRF and reported appropriately.

The investigator (or medically qualified designee) is to report all directly observed AEs and all AEs spontaneously reported by the study subject. In addition, each study subject will be questioned about AEs.

Each AE is to be assessed to determine if it meets the criteria for a SAE. If an SAE occurs, expedited reporting will follow local and international regulations, as appropriate.

When an AE occurs, it is the responsibility of the investigator (or medically qualified designee) to review all documentation (e.g., hospital progress notes, laboratory, and diagnostics reports) related to the event.

The investigator or site staff will then record all relevant information regarding an AE in the eCRF and all details relating to an SAE in the paper SAE Form provided.

It is **not** acceptable for the investigator (or medically qualified designee) to send photocopies of the subject's medical records to the sponsor in lieu of completion of the AE eCRF screen/SAE form.

There may be instances when copies of medical records for certain cases are requested by the sponsor. In this instance, all subject identifiers, except for the subject number, will be redacted on the copies of the medical records prior to submission to the sponsor.

The investigator (or medically qualified designee) will attempt to establish a diagnosis of the event based on signs, symptoms, and/or other clinical information. The diagnosis will be the documented as the AE/SAE, were known, and not the individual signs/symptoms. (e.g., upper respiratory tract infection, seasonal allergy, etc. <u>not</u> cough, runny nose).

AEs elicited by the investigator (or medically qualified designee) in a standard manner at the study visits should also be recorded in the AE section of the eCRF and/or using the SAE form (subject to the classification of the AE). Care will be taken not to introduce bias when questioning a subject about any changes in their health. Open-ended and non-leading verbal questioning should be used.

#### 10.4.1 Reporting of an Adverse Event

All AEs will be reported on the AE page of the eCRF by the investigator or site staff. It should be noted that the form for collection of SAE information is not the same as the AE eCRF screen. Where the same data are collected, the AE eCRF screen and the SAE form must be completed in a consistent manner (e.g., the same AE term should be used on both). AEs should be reported using concise medical terminology in the eCRF as well as on the paper SAE form.

#### 10.4.2 Reporting of a Serious Adverse Event

In addition to recording the details of each AE on the AE eCRF screen, an SAE form should be completed, as fully as possible. Hard copies of the paper SAE form will be provided in the investigator site master file. Original SAE forms will be retained in the investigator site master file.

Clinical Protocol

Protocol Number: 300026



It is essential to enter the following information:

- Protocol and subject identifiers
- Subject demography
- Description of events, with diagnosis (if available)
- Investigator opinion of relationship to study product (or study procedure, if appropriate)
- Criterion for seriousness.

The following are desirable and are of particular relevance for investigator and sponsor assessment of the SAE report:

- Date of onset of AE
- Date AE stopped (if relevant)
- Study product start date
- Study product end date (if relevant)
- Action taken in relation to the study product
- Outcome if known

The SAE form, completed as fully as possible, must be scanned and e-mailed to the Case Management Group mailbox PPD , with copy to the appropriate sponsor Study Manager, with the study number and subject number in the subject line of the email immediately and under no circumstance should this exceed 24 hours after study site personnel learn of the event. The investigator will submit any updated SAE data to the sponsor, immediately and under no circumstance should this exceed 24 hours of it being available.

The initial report will be followed up with more information as relevant, or as requested by the sponsor study manager. The sponsor's Study Manager will be responsible for forwarding the SAE form to other sponsor personnel as appropriate.

# 10.5 Evaluating Adverse Events

#### 10.5.1 Assessment of Intensity

The investigator or medically qualified designee will make an assessment of intensity for each AE reported during the study and will assign it to one of the following categories:

- **Mild**: An event that is easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
- **Moderate**: An event that is sufficiently discomforting to interfere with normal everyday activities
- **Severe**: An event that prevents normal everyday activities.

**NOTE**: An AE that is assessed as 'severe' should not be confused with an SAE. 'Severe' is a category utilized for rating the intensity of an event; and both non-serious AEs and SAEs can be assessed as 'severe'. For example, a headache may be 'severe' (interferes significantly with the subject's usual function) but would not be classified as 'serious' unless it met one of the criteria for SAEs, listed above. An event is defined as 'serious' when it meets at least 1 of the predefined outcomes as described in the definition of an SAE, **not** when it is rated as 'severe'.

### 10.5.2 Assessment of Causality

Clinical Protocol

Protocol Number: 300026



The causality assessment is one of the criteria used when determining regulatory reporting requirements.

For each AE (serious and non-serious), the investigator (or medically qualified designee) <u>must</u> provide an assessment of causality on the AE eCRF screen and the paper SAE form (subject to the classification of the AE). The investigator will also document in the medical notes that they have reviewed the AE and assessed causality, where applicable.

A 'reasonable possibility' of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out. Generally, the facts (evidence) or arguments to suggest a causal relationship should be provided.

The investigator will use clinical judgment to determine the relationship and will also consult the Product Information, for marketed products, in the determination of their assessment. Alternative causes, such as underlying disease(s), concomitant therapy, other risk factors, and the temporal relationship of the event to the study product will be considered and investigated.

For each AE/SAE, the investigator must document in the medical notes that they have reviewed the AE/SAE and has provided an assessment of causality.

The investigator's assessment of causality must be provided for all AEs (serious and non-serious); the investigator must record the causal relationship in the eCRF, as appropriate, and report such an assessment in accordance with the SAE reporting requirements, if applicable.

There may be situations when an SAE has occurred, and the investigator has minimal information to include in the initial report to the sponsor. However, it is very important that the investigator always make an assessment of causality for every event prior to the initial transmission of the SAE data to the sponsor. The investigator may change their opinion of causality in light of follow-up information and send an SAE follow-up report with the updated causality assessment.

# 10.6 Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow up with each subject and provide further information on the subject's condition.

All AEs (serious and non-serious) will be followed until resolution, until the condition stabilises, until the event is otherwise explained, or until the subject is lost to follow-up.

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as may be indicated or as requested by the sponsor to elucidate as fully as possible the nature and/or causality of the AE. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

New or updated information will be recorded on the AE eCRF screen and on the paper SAE form (subject to the classification of the AE).

The investigator will submit any updated SAE data to the sponsor within 24 hours of receipt of the information.

Investigators are not obliged to actively seek AEs in former subjects. However, if the investigator learns of a SAE, including death, at any time after a subject has been discharged from the study, and considers the event reasonably related to the study product or study participation, the investigator will promptly notify the sponsor by emailing the information to the Case Management Group mailbox PPD with copy to the

Property of GSK Consumer Healthcare - Confidential

Clinical Protocol

Protocol Number: 300026



appropriate sponsor Study Manager.

The investigator will submit any updated SAE data to the sponsor within the designated reporting time frames.

#### 10.7 Withdrawal Due to an Adverse Event

Withdrawal due to AEs should be distinguished from withdrawal due to other causes, according to the definition of an AE noted earlier, and recorded on the appropriate AE eCRF screen.

When a subject withdraws because of an SAE, the SAE must be reported in accordance with the reporting requirements defined.

### 10.8 Regulatory Reporting Requirements for SAEs

The sponsor has a legal responsibility to notify, as appropriate, the local regulatory authority and other regulatory authorities about the safety of a product under clinical investigation. Prompt notification of SAEs by the investigator to the sponsor is essential so that legal obligations and ethical responsibilities towards the safety of subjects are met.

The sponsor will comply with country specific regulatory requirements relating to safety reporting to the regulatory authority, Good Clinical Practice (GCP) Office/Institutional Review Board (IRB) and the investigator.

Investigator safety reports must be prepared for suspected unexpected serious adverse reactions (SUSAR) according to local regulatory requirements and sponsor policy.

An investigator who receives an investigator safety report describing a SAE or other specific safety information (e.g., summary or listing of SAEs from the sponsor) will review and then file it in the investigator site master file, and will notify the GCP office/IRB, if appropriate according to local requirements.

# 10.9 Pregnancy

# 10.9.1 Time Period for Collecting Pregnancy Information

Pregnancy information will be collected on all pregnancies reported while a female subject is participating in the study from the signing of informed consent until 5 days after last administration of study product.

#### 10.9.2 Action to be Taken if Pregnancy Occurs

The investigator will record pregnancy information on the appropriate form scan and e-mail it to the Case Management Group mailbox PPD with copy to the appropriate sponsor Study Manager. Original pregnancy information forms will be retained in the investigator site master file.

The subject will be followed to determine the outcome of the pregnancy. Information on the status of the mother and infant / neonate (including concomitant medications taken by the mother during the pregnancy) will be forwarded by the investigator to the Case Management Group mailbox PPD , with copy to the appropriate sponsor Study Manager. Generally, follow-up will be no longer than 6 to 8 weeks following the estimated delivery date. Any termination of the pregnancy will be reported.

While pregnancy itself is not considered to be an AE, abnormal pregnancy outcomes (e.g.,

Clinical Protocol

Protocol Number: 300026



spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are, and should be recorded as an SAE.

Any female subject who becomes pregnant while participating in the study will be withdrawn.

#### 11 DATA MANAGEMENT

As used in this protocol, the term CRF is understood to refer to either a paper form or an electronic data record or both, depending on the data collection method.

For this study, subject data will be entered into an electronic CRF (eCRF), using a validated system. Data relating to clinical screening/efficacy assessments, SAEs and pregnancy will also be collected on paper forms.

The investigator is responsible for verifying that data entries are accurate and correct by physically or electronically signing the CRF.

The source documents (e.g. hospital records, clinical and office charts, laboratory notes, memoranda, subject diaries, questionnaires, evaluation checklists, pharmacy dispensing records, recorded data from automated instruments, microfiches, photographic negatives, microfilm or magnetic media, x-rays, subject files and records kept at the pharmacy, at the laboratory and at the medico-technical departments involved in the clinical study) which contain the source of data recorded in the eCRF should be specified. The eCRF, paper forms and diary can be used as a source document at the discretion of data management.

Each subject will be assigned and identified by a unique Screening Subject Number. Any reference made to an individual subject within the study must be done using their unique Screening Subject Number.

# 11.1 Case Report Form

A CRF is a printed, optical, or electronic document designed to record the protocol required information to be reported to the sponsor on each trial subject. For each subject who has given informed consent/assent, the eCRF must be completed and signed by the investigator (or authorized designee) to certify the data are complete and correct. The investigator must maintain accurate documentation (source data) that supports the information entered in the eCRF.

Management of clinical data will be performed in accordance with Third Party Biostatistics and Data Management (BDM) Vendor applicable standards and data cleaning procedures with oversight by the sponsor to ensure integrity of the data, for example, to remove errors and inconsistencies in the data.

To protect the privacy of subjects, no Personal Information (PI) (including the subject's name or initials or full birth date) is to be recorded in the eCRF or as part of the query text.

All eCRF pages should be completed during a subject assessment when the eCRF has been designated as the source. Data that is sourced elsewhere should be entered into the eCRF in an agreed upon timeframe between the investigator and sponsor.

The sponsor will obtain and retain all eCRFs and associated study data as applicable at the completion of the study.

Clinical Protocol

Protocol Number: 300026



# 11.2 Data Handling

Documentation of all data management activities should allow step-by-step retrospective assessment of data quality and study performance.

Any changes or corrections to data will be performed in the Electronic Data Capture (EDC) System, which will include rationale for changes. The EDC system has an audit trail, which will provide a complete record of the changes and corrections endorsed by the investigator.

AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) and any concomitant medication terms (if applicable) using a validated medication dictionary, WHODrug.

#### 11.2.1 Data Queries

Programmed edit checks will be generated automatically, as the data are being entered into the system. Reports and listings on the eCRF data will also be run, in addition to the queries already programmed and generated by the system, to raise manual queries as needed for site clarification or correction. The third-party vendor will raise queries as needed on safety data to code the terms (AEs and Drugs or concomitant medication) appropriately.

The study monitor will perform ongoing review the of the eCRFs in accordance with the monitoring plan, to confirm that data entered into the eCRF by authorised site personnel are accurate, complete, and verifiable from source documents; that the safety and rights of participants are being protected; and that the study is being conducted in accordance with the currently approved protocol and any other study agreements, ICH GCP, and all applicable regulatory requirements.

Any queries will be generated in the EDC System to the investigator or designee, enabling the errors to be addressed in parallel with Data Management review. The monitor can also run reports and listings on the eCRFs to raise manual queries, as needed, for site clarification or correction.

# 12 STATISTICAL CONSIDERATIONS AND DATA ANALYSES

# 12.1 Sample Size Determination

Sufficient subjects will be screened to randomize approximately 240 subjects to study treatment to ensure approximately 235 complete the study (approximately 94 subjects each for test toothpaste and negative control, and 47 subjects for positive control), allowing for 2% dropouts after randomization, as observed in previous clinical studies conducted in China.

The study will be powered sufficiently to demonstrate statistical superiority of the test toothpaste compared to the negative control for the change from Baseline in the Schiff sensitivity score after 12 weeks of treatment.

The true effect size is expected to be 0.5 (effect size (ES) = mean difference [test toothpaste – negative control] / pooled standard deviation [SD]; mean difference = 0.3, SD=0.6). Such assumptions would also infer at least a 15% superior relative mean change from Baseline for the test toothpaste compared to the negative control (assuming mean change from a Baseline Schiff sensitivity score for negative control less than 2), a requirement of the Chinese MoH guidelines for the testing of functional (desensitising) toothpastes for at least one clinical DH measure (Ministry of Health (China), 2010).

Clinical Protocol

Protocol Number: 300026



With 94 subjects per group (for test toothpaste and negative control arms), there is 92.65% power to detect an effect size of 0.5 at the two-sided 5% significance level based on a two-sample t-test (using PASS software version 19.0.1).

Estimates of the above dropout rate and SD are based on results from three similar clinical studies (sponsor clinical studies: 205794, 208153, 216954).

The positive control has clinically proven longer-term DH efficacy in two clinical studies conducted in China on Chinese populations (sponsor clinical studies: which satisfied the China MoH requirements (Ministry of Health (China), 2010). As such, it has been included in this study as a benchmark of performance in the Chinese population for 'study validation'; 47 subjects in the positive control group are deemed sufficient to demonstrate statistical superiority for positive vs. negative controls.

# 12.2 Populations for Analysis

#### 12.2.1 Definitions of Analysis Populations

The Safety population will include all randomized subjects who complete at least one use of study product. This population will be based on the study product the subject received. All assessments of safety will be based on this analysis population.

The modified Intent-To-Treat (mITT) population will include all randomized subjects who complete at least one use of study product and have at least one post Baseline efficacy assessment. This population will be based on the study product to which the subject was randomized. All assessments of efficacy will be primarily based on this analysis population.

The per protocol (PP) population is defined as all subjects in the mITT population who have at least one assessment of efficacy considered unaffected by protocol deviations.

# 12.2.2 Exclusion of Data from Analysis

Exclusion of any data from the analyses will be determined during Blinded Data Review (BDR) prior to database lock. Any reasons for exclusion from an analysis population will be listed, if applicable.

A PP analysis will be performed for each change from Baseline in Schiff sensitivity score and tactile threshold endpoints if there is more than 10% difference in the number of subjects between the PP and mITT populations. A decision to perform a PP analysis should be made prior to study unblinding (release of the randomization codes).

# 12.3 Statistical Analyses

This is a summary of the planned statistical analyses; the detail of the proposed statistical analyses will be documented in the statistical analysis plan (SAP), written following finalization of the protocol and prior to study unblinding.

Significance testing will be conducted at the two-sided 5% significance level.

Schiff sensitivity score, tactile threshold (g) and VAS (mm) will be derived as the average score or value, respectively, of the 2 test teeth (identified at Baseline). Change from Baseline will be derived for the individual teeth first before calculating the average change of the 2 test teeth.

Clinical Protocol

Protocol Number: 300026



#### 12.3.1 Primary Analysis

The primary endpoint of this study is the change from Baseline in the Schiff sensitivity score at Week 12; the primary hypothesis test will be the comparison between the test toothpaste and the negative control in the mITT population.

Change from Baseline in Schiff sensitivity score will be analysed using a Mixed Model with Repeated Measures (MMRM), with study product, visit and study product by visit interaction as fixed effects, and Baseline Schiff sensitivity score as a covariate. Subject will be included as a repeated measure with unstructured covariance matrix. Kenward Rogers degrees of freedom approach will be applied (Kenward and Roger, 1997). The difference between least square means for the test toothpaste compared to the negative control at Week 12 will be presented along with two-sided p-value and 95% CIs.

As a sensitivity analysis, the change from Baseline in Schiff sensitivity score at Week 12 will be compared between study products (test toothpaste vs. negative control) using an Analysis of Covariance (ANCOVA) model with study product as a fixed effect and Baseline Schiff sensitivity score as a covariate.

The assumption of normality and homogeneity of variance in each MMRM will be investigated. In case of violation of these assumptions, a suitable non-parametric test (adjusted for the randomisation stratification) will be performed to assess change from Baseline comparisons (test toothpaste vs. negative control at Week 12) and the results will be provided to support the MMRM results; the non-parametric results will be considered confirmatory under the observation of strong violations of the assumptions.

### 12.3.2 Secondary Analyses

Change from Baseline in Tactile Threshold (g) at Week 12:

Change from Baseline in tactile threshold (g) will be analysed using the same MMRM as the primary endpoint but with Baseline tactile threshold (g) as a covariate, rather than Baseline Schiff sensitivity score. In addition, the maximum Baseline Schiff sensitivity score of the two test teeth (2 or 3) will be fitted as a fixed effect. The difference between least square means for the test toothpaste vs. negative control at Week 12 will be presented, along with the two-sided p-value and 95% CIs.

As a sensitivity analysis, the change from Baseline in tactile threshold (g) at Week 12 will be compared between study products (test toothpaste vs. negative control) using an Analysis of Covariance (ANCOVA) model with study product and the maximum Baseline Schiff sensitivity score of the two test teeth (2 or 3) as fixed effects and the Baseline tactile threshold (g) as a covariate.

#### Change from Baseline in VAS (mm) at Week 12:

Change from Baseline in VAS (mm) will be analysed using the same MMRM and ANCOVA (as a sensitivity analysis) as for the change from Baseline in tactile threshold (g) but with Baseline VAS (mm) as a covariate, rather than the Baseline tactile threshold (g). The difference between least square means for the test toothpaste vs. negative control at Week 12 will be presented, along with the two-sided p-value and 95% CIs.

Clinical Protocol

Protocol Number: 300026



#### Other Secondary Endpoints:

- Test toothpaste vs. negative control
  - Change from Baseline in Schiff sensitivity score, tactile threshold (g) and VAS (mm) at Week 6
- Positive control vs. negative control
  - Change from Baseline in Schiff sensitivity score, tactile threshold (g) and VAS (mm) at Week 6 and Week 12.

These other secondary endpoint analyses will utilise the results at Week 6 (test toothpaste vs. negative control and positive vs. negative control) and Week 12 (positive vs. negative control) from the same respective MMRM model applied for the change from Baseline in Schiff sensitivity score, tactile threshold (g) and VAS (mm) described above.

The results from each MMRM will be tabulated together, presenting the following information, in addition to the results already specified for the primary and secondary analyses above.

- Least square mean change from Baseline for each study product at Week 6 and Week 12 (based on the observed stratification margins for tactile threshold model) and used to test for any change from Baseline with two-sided p-values and 95% CIs.
- Differences between least square mean change from Baseline (test toothpaste vs. negative control at Week 6, positive control vs. negative control at Week 6 and Week 12) with two-sided p-values and 95% CIs.

The assumption of normality and homogeneity of variance in each MMRM will be investigated. In case of violation of these assumptions, a suitable non-parametric test (adjusted for the randomisation stratification) will be performed for each required secondary endpoint comparison between study products at each time point and results will be provided to support the MMRM results; the non-parametric results will be considered to supersede the MMRM results under the observation of strong violations of the assumptions.

The ANCOVA sensitivity analysis results at Week 12 for positive vs. negative control for each endpoint will be obtained from the same ANCOVA models using Week 12 data as described above for the test toothpaste vs. negative control comparisons. As additional sensitivity analyses, the change from Baseline in Schiff sensitivity score, tactile threshold (g) and VAS (mm) at Week 6 will be analysed using the same ANCOVA model as for the Week 12 sensitivity analyses detailed above.

#### 12.3.3 Safety Analyses

Safety analyses will be performed on the Safety population, according to study product received. AEs will be regarded as 'treatment emergent' if they occur on or after the first study product use at Baseline (Visit 1). In case of misallocation, compared to the randomisation schedule, TEAEs will be associated with the most recent study product received.

Each AE will be categorized as oral or non-oral by the investigator, or medically qualified designee. All will be reviewed by the CRS prior to database lock and unblinding, and coded using the MedDRA.

A listing of all AEs will be presented for all subjects in the Safety population with the following AEs summaries (number of distinct AEs and frequency/proportion of subjects affected) will be presented by product group and overall:

Clinical Protocol

Protocol Number: 300026



- Treatment emergent AEs
- Treatment emergent AEs by System Organ Class (SOC) and Preferred Term (PT)
- Treatment emergent AEs by Oral/Non-Oral and PT
- Treatment emergent treatment related AEs by Oral/Non-Oral and PT
- Treatment emergent treatment related serious AEs by SOC and PT

Separate listings will be presented for:

- Deaths, SAEs and any AEs leading to product or study discontinuation.
- OST findings (with a summary of abnormalities by visit)
- OHT findings (with a summary of changes by visit)
- Exposure to study product <u>Section 12.3.5.1.</u>

#### 12.3.4 Demographic and Baseline Characteristics

Demographic and Baseline characteristics will be summarized by treatment group for the Safety and mITT populations, and the PP population if a PP analysis is performed.

Categorical variables (such as sex, race and Baseline Schiff stratification score) will be summarized by the number and percentage of subjects with each relevant characteristic in each product group. Continuous variables such as (age) will be summarized by mean, SD, median, minimum and maximum values in each product group.

# 12.3.5 Study Product Compliance and Use of Other Therapies

#### 12.3.5.1 Study Product Compliance

Compliance with product use (number of brushings) will be listed and summarized for the mITT population at each visit, and cumulatively for the overall treatment period (for most subjects this will be 12 weeks) by product group.

Number of expected brushings =  $2 \times \text{Number of days between Visit X and Visit (X+1)}$ 

Number of actual brushings = (Number of expected brushings) - (Number of missed

brushings) + (Number of additional brushings)

% Compliance at 'Visit X' = (Number of actual brushings prior to Visit X)  $\times 100$ 

(Number of expected brushings prior to Visit X)

#### 12.3.5.2 Prior and Concomitant Medications and Treatments

Prior medications, concomitant medications and significant non-drug therapies taken during the study will be listed for the Safety population.

#### 12.3.6 Handling of Dropouts and Missing Data

MMRM analyses account for missing data using 'a missing at random' assumption, i.e., there is a systematic relationship between the propensity for missing values and the observed data, but not the missing data. Under such assumptions, MMRM is shown to provide unbiased estimates of the treatment effect, whilst the analysis of only complete cases using ANCOVA are biased (Baron et al., 2008; Ashbeck et al., 2016). Such complete case analysis requires a 'missing completely at random' assumption to remain unbiased and this is unlikely to hold, i.e., the fact that the data are missing is independent of the observed and unobserved data.

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH

Clinical Protocol

Protocol Number: 300026



Using an MMRM, it will therefore be assumed that a subject with missing data at one post-Baseline visit would have obtained a similar efficacy result at that visit compared to a subject using the same study product with similar non-missing results at other timepoints (Baseline and the other post-Baseline visit).

Sensitivity analyses will present results from the separate ANCOVA models using only non-missing values at each single time point. Additional sensitivity analyses may be added to the SAP prior to unblinding in case of high drop-out rates and/or exclusion from PP population.

#### 12.3.7 Interim Analysis

No interim analysis is planned for this study

#### 13 STUDY GOVERNANCE CONSIDERATIONS

# 13.1 Quality Control

In accordance with applicable regulations, including GCP and the sponsor's procedures, the sponsor or designee (i.e., third-party vendor monitors) will contact the site to review the protocol, study requirements, and staff responsibilities with study personnel prior to the start of the study to satisfy regulatory, ethical, and sponsor requirements. When reviewing data collection procedures, the discussion will include identification, agreement and documentation of data items for which the eCRF will serve as the source document.

The sponsor or designee will monitor the study and site activity to verify:

- Data are authentic, accurate, and complete.
- Safety and rights of subjects are being protected.
- Study is conducted in accordance with the currently approved protocol and any other study agreements, GCP, and all applicable regulatory requirements.

The extent and nature of monitoring will be described in a written monitoring plan on file at the sponsor. The investigator (or designee) agrees to allow the monitor(s) direct access to all relevant documents and agrees to co-operate with the monitor(s) to ensure that any problems detected during these monitoring visits are resolved.

# 13.2 Quality Assurance

To ensure compliance with GCP and all applicable regulatory requirements, the sponsor may conduct a quality assurance assessment and/or audit of the site records, and regulatory agencies may conduct regulatory inspections at any time during or after completion of the study.

In the event of an assessment, audit or inspection, the investigator (and institution) must agree to grant the advisor(s), auditor(s) and inspector(s) direct access to all relevant documents and to allocate their time and the time of their staff to discuss the conduct of the study, any findings/relevant issues and to implement any corrective and/or preventative actions to address any findings/issues identified.

The investigator will notify the sponsor or its agents immediately of any regulatory inspection notification in relation to the study. Furthermore, the investigator will cooperate with the sponsor or its agents to prepare the study site for the inspection and will allow GSK CH or its agent, whenever feasible, to be present during the inspection. The investigator will promptly supply copies of the inspection finding to the sponsor or its agent. Before response submission

Clinical Protocol

Protocol Number: 300026



to the regulatory authority, the investigator will provide the sponsor or its agents with an opportunity to review and comment on responses to any findings.

The sponsor will be available to help the investigator prepare for an inspection.

#### 13.3 **Regulatory and Ethical Considerations**

#### 13.3.1 Institutional Review Board

It is the responsibility of the investigator to have prospective approval of the study protocol, protocol amendments, informed consent documents, investigator brochure/safety statement (including any updates) and other relevant documents (e.g., recruitment advertisements, if applicable) from the GCP Office/IRB. All correspondence with the GCP Office/IRB should be retained in the investigator site file. Copies of GCP Office/IRB approvals should be forwarded to the sponsor prior to the initiation of the study, and also when amendments to the protocol are made.

The only circumstance in which an amendment may be initiated prior to GCP Office/IRB approval is where the change is necessary to eliminate apparent immediate hazards to the subjects. In that event, the investigator must notify the GCP Office/IRB and sponsor in writing immediately after the implementation.

#### 13.3.2 **Ethical Conduct of the Study**

The study will be conducted in accordance with the protocol and legal and regulatory requirements, as well as the general principles set forth in the International Ethical Guidelines for Biomedical Research Involving Human Subjects (Council for International Organizations of Medical Sciences 2002), International Ethical Guidelines for Health-Related Research Involving Humans (Council for International Organizations of Medical Sciences, 2016), guidelines for GCP (ICH 1996 and revision 2), and the Declaration of Helsinki (World Medical Association 2013).

In addition, the study will be conducted in accordance with the protocol, the ICH guideline on GCP, and applicable local regulatory requirements and laws.

#### 13.3.3 **Subject Information and Consent**

All parties will ensure protection of subject personal data and will not include subject names or other identifiable data in any reports, publications, or other disclosures, except where required by laws.

When study data are compiled for transfer to the sponsor and other authorised parties, subject names, addresses, and other identifiable data will be replaced by numerical codes based on a numbering system provided by the sponsor in order to de-identify study subjects.

Note that the use of initials should be avoided.

The study site will maintain a confidential list of subjects who participated in the study, linking each subject's numerical code to his or her actual identity. In case of data transfer, the sponsor will maintain high standards of confidentiality and protection of subjects' personal data consistent with applicable privacy laws.

The informed consent document must be in compliance with ICH GCP, local regulatory requirements, and legal requirements, including applicable privacy laws.

Clinical Protocol

Protocol Number: 300026



The informed consent document used during the informed consent process must be reviewed and approved by the sponsor, approved by the GCP Office/IRB before use, and available for inspection.

The investigator must ensure that each study subject, is fully informed about the nature and objectives of the study and possible risks associated with participation.

# 13.3.4 Subject Recruitment

Advertisements approved by GCP Office/IRB and investigator databases may be used to recruit study subjects. Use of a GCP Office/IRB approved, generic, pre-screening questionnaire to determine general eligibility for this study is allowed. This pre-screening questionnaire may be used by sites as a phone script and/or to review internal databases to identify subjects. The sponsor will have an opportunity to review and approve the content of any study recruitment materials directed to potential study subjects before such materials are used.

# 13.3.5 Reporting of Safety Issues and Serious Breaches of the Protocol or ICH GCP

The investigator will inform the sponsor immediately of any urgent safety measures taken by the investigator to protect the study subjects against any immediate hazard, and of any serious breaches of this protocol or of ICH GCP the investigator becomes aware of.

The sponsor defines a serious breach as a breach likely to affect to a significant degree the safety and rights of a subject or the reliability and robustness of the data generated in sponsored human subject research studies.

In the event of any prohibition or restriction imposed (i.e., clinical hold) or if the investigator is aware of any new information that might influence the evaluation of the benefits and risks of the investigational product, the sponsor should be informed immediately.

# 13.4 Posting of Information on Publicly Available Clinical Trial Registers

Study-related information from this protocol will be posted on publicly available clinical trial registers before enrollment of subjects begins in accordance with applicable sponsor's processes. The sponsor intends to make anonymized subject-level data from this trial available to external researchers for scientific analyses or to conduct further research that can help advance medical science or improve patient care. This helps ensure the data provided by trial participants are used to maximum effect in the creation of knowledge and understanding.

# 13.5 Provision of Study Results to Investigators

Where required by applicable regulatory requirements, an investigator signatory will be identified for the approval of the clinical study report. The investigator will be provided reasonable access to statistical tables, figures and relevant reports, and will have the opportunity to review the complete study results. The sponsor will also provide the investigator with the full summary of the study results. The investigator is encouraged to share the summary results with the study subjects, as appropriate.

A manuscript will be progressed for publication in the scientific literature if the results provide important scientific or medical knowledge. The procedures and timing for public disclosure of the results summary and for development of a manuscript for publication will be in accordance with the sponsor's policy.

Property of GSK Consumer Healthcare - Confidential

May not be used, divulged, published or otherwise disclosed without the consent of GSKCH

Clinical Protocol

Protocol Number: 300026



#### 13.6 Records Retention

Following closure of the study, the investigator must maintain all site study records (except for those required by local regulations to be maintained elsewhere), in a safe and secure location.

The records (study/ site master file) must be maintained to allow easy and timely retrieval, when needed (e.g., for a sponsor audit or regulatory inspection) and must be available for review in conjunction with assessment of the facility, supporting systems, and relevant site staff.

Where permitted by local laws/regulations or institutional policy, some or all of these records can be maintained in a format other than hard copy (e.g., microfiche, scanned, electronic); however, caution needs to be exercised before such action is taken.

The investigator must ensure that all reproductions are legible and are a true and accurate copy of the original and meet accessibility and retrieval standards, including re-generating a hard copy, if required. Furthermore, the investigator must ensure there is an acceptable back-up of these reproductions and that an acceptable quality control process exists for making these reproductions.

The investigator must assure that the subject's anonymity will be maintained. On CRFs or other documents submitted to the sponsor, subjects should not be identified by their names or initials, but by an identification code. The investigator should keep a separate log of subjects' codes, names and addresses. Documents not for submission to the sponsor (e.g., subjects' written consent forms) should be maintained by the investigator in strict confidence.

Records and documents, including signed ICF, pertaining to the conduct of this study must be retained by the investigator as per the signed contractual agreement, from the issue of the final Clinical Study Report (CSR) or equivalent summary, unless local regulations or institutional policies require a longer retention period. The minimum retention time will meet the strictest standard applicable to that site for the study, as dictated by any institutional requirements or local laws or regulations, sponsor standards/procedures, and/or institutional requirements.

No study document should be destroyed without a prior written agreement between the sponsor and the investigator. The investigator must notify the sponsor of any changes in the archival arrangements, including, but not limited to, archival at an off-site facility or transfer of ownership of the records in the event the investigator is no longer associated with the site.

# 13.7 Conditions for Terminating the Study

Premature termination of this study may occur because of a regulatory authority decision, change in opinion of the GCP Office/IRB, or study product safety problems, or at the discretion of the sponsor.

If a study is prematurely terminated, the sponsor will promptly notify the investigator. After notification, the investigator must promptly contact all participating subjects and should assure appropriate therapy/ follow-up for the subjects. As directed by the sponsor, all study materials must be collected and all CRF's completed to the greatest extent possible. Where required by the applicable regulatory requirements, the sponsor should inform the regulatory authority(ies) and the investigator should promptly inform the GCP Office/IRB and provide the GCP Office/IRB with a detailed written explanation of the termination or suspension.

If the GCP Office/IRB terminates or suspends its approval/favorable opinion of a trial, the investigator should promptly notify the sponsor and provide the sponsor with a detailed written explanation of the termination or suspension.

Clinical Protocol

Protocol Number: 300026



Upon completion or premature discontinuation of the study, the sponsor's monitor will conduct site closure activities with the investigator or site staff, as appropriate, in accordance with applicable regulations including GCP, and the sponsor's Standard Operating Procedures.

#### 14 REFERENCES

Addy M. Dentine hypersensitivity: Definition, prevalence, distribution and aetiology. Tooth wear and sensitivity. 2000, 239-48.

Addy M. Dentine hypersensitivity: New perspectives on an old problem. International Dental Journal. **2002**, *52*, 367-375.

Addy M., Mostafa P., Absi E., Adams D. Cervical dentin hypersensitivity. Etiology and management with particular reference to dentifrice. In *Proceedings of Symposium on Hypersensitive Dentin. Origin and Management*; Rowe, N., Ed.; University of Michigan, Ann Arbor, MI, 1985; 147–167.

Aghazadeh Z., Behroozian A., Najafi H., Faramarzi M. Comparison of gingival and dental indices in lactating and non-lactating mothers during first 6 month after delivery. *Pesqui Bras Odontopediatria Clin Integr* 2019; 19:e4586

Ashbeck E.L., Bell M.L. Single time point comparisons in longitudinal randomized controlled trials: power and bias in the presence of missing data. *BMC Med Res Methodol*, 2016, 16, 43.

Baron G., Ravaud P., Samson A., et al. Missing data in randomized controlled trials of rheumatoid arthritis with radiographic outcomes: A simulation study. Arthritis Rheum-Arthritis Care Res. 2008;59:25–31

Brännström M., A hydrodynamic mechanism in the transmission of pain producing stimuli through dentin. In *Sensory Mechanisms in Dentin*; Anderson, D., Ed.; Oxford: Pergamon Press, 1962; 73–79.

Canadian Advisory Board on Dentin Hypersensitivity, Consensus-based recommendations for the diagnosis and management of dentin hypersensitivity. *J. Can. Dent. Assoc.* **2003**, *69*, 221–226.

Dempsey Pa, Townsend G. Genetic and environmental contributions to variation in human tooth size. Heredity. 2001;86(6):685.

Docimo R., Montesani L., Maturo P., Costacurta M., Bartolino M., Zhang Y. P., DeVizio W., Delgado E., Cummins D., Dibart S., et al., Comparing the efficacy in reducing dentin hypersensitivity of a new toothpaste containing 8.0% arginine, calcium carbonate, and 1450 ppm fluoride to a benchmark commercial desensitizing toothpaste containing 2% potassium ion: An eight-week clinical study . *J. Clin. Dent.* **2009**, *20*, 137–143.

Fischer C., Fischer R. G., Wennberg A., Prevalence and distribution of cervical dentine hypersensitivity in a population in Rio de Janeiro, Brazil. *J. Dent.* **1992**, *20*, 272–276.

Flynn J., Galloway R., Orchardson R., The incidence of "hypersensitive" teeth in the West of Scotland. *J. Dent.* **1985**, *13*, 230–236.

Hall R., Embery G., Shellis R., Biological and structural features of enamel and dentin: current concepts relevant to erosion and dentin hypersensitivity. In *Tooth Wear and Sensitivity*; Addy, M., Embery, G., Edgar, W., Orchardson, R., Eds.; Martin Dunitz Ltd, London, **2000**; pp 3–19.

Hall C., Mason S., Cooke J. Exploratory randomised controlled clinical study to evaluate the

Page 66 of 73

Clinical Protocol

Protocol Number: 300026



comparative efficacy of two occluding toothpastes—a 5% calcium sodium phosphosilicate toothpaste and an 8% arginine/calcium carbonate toothpaste—for the longer-term relief of dentine hypersensitivity. *J Dent.* **2017**, 60, 36-42.

Holland G. R., Narhi M. N., Addy M., Gangarosa L., Orchardson R., Guidelines for the design and conduct of clinical trials on dentine hypersensitivity. *J. Clin. Periodontol.* **1997**, *24*, 808–813.

#### ICH E6 (R2) Good clinical practice | European Medicines Agency (europa.eu)

K Kenward M.G., Roger J. Small sample inference for fixed effects from restricted maximum likelihood. Biometrics. **1997**, 983-997.

Laster L., Laudenbach K. W., Stoller N. H., An evaluation of clinical tooth mobility measurements. *J. Periodontol.* **1975**, *46*, 603–607.

Leight R., Bowman J., Barlow A., Dentinal Hypersensitivity: Evidence for a "No Treatment" Effect. J. Dent. Res. **2008**, 87, Abstract No 3498.

Liang X, Wei Z, Hu D, *et al.* Prevalence of dentin hypersensitivity among the residents of xi'an city, china. Acta Odontologica Scandinavica. **2017**;75(6):387-93.

Lobene R. R., Weatherford T., Ross N. M., Lamm R. A., Menaker L., A modified gingival index for use in clinical trials. *Clin. Prev. Dent.* **1986**, *8*, 3–6.

Makin S. A., Stannous fluoride dentifrices. Am. J. Dent. 2013, 26 Spec No. 3A – 9A.

Ministry of Health, China. Efficacy evaluation of toothpaste - Part 4: Guidelines for efficacy evaluation on dentin hypersensitivity. Health Industrial Standard of the People's Republic of China. WS/T 326.4-2010.

Ni, L.X., He, T., Chang, A. and Sun, L., 2010. The desensitizing efficacy of a novel stannous-containing sodium fluoride dentifrice: An 8-week randomized and controlled clinical trial. *American Journal of Dentistry*, 23, p.17B.

Orchardson R., Gillam D.G., The efficacy of potassium salts as agents for treating dentin hypersensitivity. *J. Orofac. Pain*, **2000**, *14*, 9-19.

Parkinson CR and R Willson. A comparative in vitro study investigating the occlusion and mineralization properties of commercial dentifrices in a four day dentine disc model. J. Clin. Dent. Spec Issue, 22(3) 2011.

Parkinson C, Hughes N, Jeffery P, *et al.* The efficacy of an experimental dentifrice containing 0.454% w/w stannous fluoride in providing relief from the pain of dentin hypersensitivity: An 8-week clinical study. American journal of dentistry. 2013;26:25A-31A.

Parkinson C, Hughes N, Targett D, Ferrier A, Jones S B, Seong J, Davies M, Macdonald E L, West N. Dentine tubule occlusion of an experimental anti-sensitivity toothpaste in-situ. IADR 2013.

Parkinson CR, Jeffery P, Milleman JL, *et al.* Confirmation of efficacy in providing relief from the pain of dentin hypersensitivity of an anhydrous dentifrice containing 0.454% with or without stannous fluoride in an 8-week randomized clinical trial. American journal of dentistry. 2015;28(4):190-6.

Pashley D. H., Dentin permeability, dentin sensitivity, and treatment through tubule occlusion, J Endodont. 1986, 12, 465-474.

Clinical Protocol

Protocol Number: 300026



Pashley D., Tay F., Haywood V., Collins M., Drisko C., Consensus-based recommendations for the diagnosis and management of dentin hypersensitivity. *Compend Cont Edu Dent* **2008**, *29*, 1–35.

Polson A, Caton J, Yeaple R, *et al.* Histological determination of probe tip penetration into gingival sulcus of humans using an electronic pressure - sensitive probe. Journal of Clinical Periodontology. 1980;7(6):479-88.

Rees J. S., The prevalence of dentine hypersensitivity in general dental practice in the UK. *J. Clin. Periodontol.* **2000**, *27*, 860–865.

#### Rulemaking History for OTC Oral Healthcare Drug Products | FDA

Samant A, Malik C, Chabra S, et al. Gingivitis and periodontal disease in pregnancy. Journal of Periodontology. 1976, 47(7): 415-8.

Schiff T, Dotson M, Cohen S, *et al.* Efficacy of a dentifrice containing potassium nitrate, soluble pyrophosphate, pvm/ma copolymer, and sodium fluoride on dentinal hypersensitivity: A twelve-week clinical study. The Journal of clinical dentistry. 1994;5:87-92.

Schiff T., He T., Sagel L., Baker R., Efficacy and safety of a novel stabilized stannous fluoride and sodium hexametaphosphate dentifrice for dentinal hypersensitivity. *J. Contemp. Dent. Pract.* **2006**, *7*, 1–8.

Seltzer S., Bender I., *The Dental Pulp: Biologic Considerations in Dental Procedures*; JP Lippincott, 1975.

Sponsor Clinical Study 205794, A study to evaluate the efficacy of an experimental occlusion technology dentifrice in the relief of dentinal hypersensitivity. GSK data held on file; 2017-



# CCI

Sponsor Clinical Study 216953. A Real-world Evidence Study Evaluating Oral Health Related Quality Of Life Following The Use Of Antisensitivity Toothpaste For Dentine Hypersensitivity Management. GSK data held on file; 2022

Sponsor Clinical Study 216954. An 8 Week, Randomised, Examiner-blind, Controlled Clinical Study to Evaluate the Efficacy of a Stannous Fluoride Dentifrice in the Relief of Dentinal Hypersensitivity in a Chinese Population. GSK data held on file; 2022.

Sponsor Clinical Study 208153. A Randomized, 8 Week Clinical Study to Evaluate the Efficacy of an Experimental Stannous Fluoride Dentifrice in the Relief of Dentinal Hypersensitivity. GSK data held on file; 2018.

West N. X., Addy M., Jackson R. J., Ridge D. B., Dentine hypersensitivity and the placebo response. A comparison of the effect of strontium acetate, potassium nitrate and fluoride toothpastes. J. Clin. Periodontol. 1997, 24, 209–215.

World Medical Association Declaration of Helsinki, 64th General Assembly, Fortaleza 2013.

Protocol Number: 300026



# 15 APPENDICES

#### 15.1 ABBREVIATIONS

The following is a list of abbreviations that may be used in the protocol.

Table 15-1 Abbreviations

| Abbreviation | Term |
|------------------|-------------------------------------------|
| AE | Adverse event |
| ANCOVA | Analysis of Covariance |
| BDM | Biostatistics and Data Management |
| BDR | Blinded data review |
| CI | Confidence interval |
| CRF | Case report form |
| CRS | Clinical Research Scientist |
| CSPS | calcium sodium phosphosilicate |
| DH | Dentine hypersensitivity |
| EAR | Erosion, Abrasion, Recession |
| ECs | Ethics committees |
| EDC | Electronic data capture |
| ECG | Electrocardiogram |
| eCRF | Electronic case report form |
| ES | Effect size |
| g | Gram |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| ICH | International Conference on Harmonisation |
| IRB | Institutional Review Board |
| IRT | Interactive Response Technology |
| OHT | Oral hard tissue |
| OST | Oral soft tissue |
| OTC | Over-the-counter |
| MFC | Manufacturing formulation code |
| MGI | Modified gingival index |
| mITT | Modified Intent to Treat |
| MMRM | Mixed model with repeated measures |
| МОН | Ministry of Health |
| NaF | Sodium fluoride |
| N/A | Not applicable |
| PI | Personal information |
| PP | Per protocol |
| P&G | Proctor and Gamble |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SnF <sub>2</sub> | Stannous fluoride |

Property of GSK Consumer Healthcare - Confidential

# 300026 Protocol Amendment Project Ox 14 Feb 2023 | TMF-238226 | 3.0

GSK Consumer Healthcare Clinical Protocol

Protocol Number: 300026



| Abbreviation | Term |
|--------------|-----------------------------------------------|
| SUSAR | Suspected unexpected serious adverse reaction |
| TEAEs | Treatment emergent adverse events |
| UK | United Kingdom |
| US | United States |
| VS | Versus |

Protocol Number: 300026



# 15.2 Screening questionnaire

1. Which of the following best describe any sensations that you may have felt in your teeth? (tick all that apply)

| Itchy | Aching | Shooting |
|-------------|---------------|------------|
| Piercing | Tingling | Sharp |
| Dull | Flashing | Shivery |
| Lingering | Twinging | Flickering |
| Stabbing | Shattering | Freezing |
| Fleeting | Quivering | Pricking |
| Pain | Discomfort | Twinges |
| Sensitivity | None of these | |

If answer is 'None of these', EXCLUDE

From now on we are going to call what you feel, the 'sensations in your teeth' or 'sensations'.

2. How long have you been experiencing any sensations in your teeth? (tick only one response)

| Less than six months | Exclude |
|---------------------------------------------|---------|
| More than six months but less than a year | Proceed |
| More than a year but less than five years | Proceed |
| More than five years but less than 10 years | Proceed |
| More than 10 years | Exclude |
| None | Exclude |

3. Which parts of your mouth have been affected by these sensations? (tick all that apply)

| Top front | Proceed |
|--------------|---------|
| Top back | Proceed |
| Bottom front | Proceed |
| Bottom back | Proceed |
| None | Exclude |

Protocol Number: 300026



4. Which of the following cause you to have sensations in your teeth? (tick all that apply)

| Cold fluids | Acidy fruits (e.g., oranges) | Having teeth cleaned at the dentist |
|---|---|---|
| Hot foods | Sweet things | Tooth Whitening Products |
| Hard foods | Sticky foods | Metals touching my teeth |
| Cold air | Ice Cream | flossing certain teeth |
| Salty foods | Cold foods | Tooth brushing |
| Hot fluids | None of these | |

If answer is 'None of these', EXCLUDE

5. How often do you experience these sensations in your teeth?

| Several times a day | Proceed |
|------------------------|---------|
| Once a day | Proceed |
| Several times a week | Proceed |
| Once a week | Proceed |
| Several times a month | Exclude |
| Once a month | Exclude |
| Less than once a month | Exclude |
| Never | Exclude |

6. If you have any sensations, on average how long do these sensations last? (tick only one response)

| A few seconds | Proceed |
|--------------------------|---------|
| About a minute | Proceed |
| Several minutes | Proceed |
| About half an hour | Proceed |
| Longer than half an hour | Exclude |
| Don't have them | Exclude |

Protocol Number: 300026



# 15.3 Video Compliance Check-list

| Did the subject only use the study products provided? | Yes | No* |
|---|---|---|
| Did the subject use the correct amount of toothpaste (full toothbrush head)? | Yes | No* |
| Did the subject brush according to the acclimatisation product usage instructions? | Yes | No* |
| Did the subject rinse with water during tooth brushing? | Yes** | No |
| Did the subject rinse with the correct amount of water after brushing? | Yes | No* |
| If the subject brushed their tongue, did they do this after toothbrushing? N/A (circle if subject did not brush their tongue) | Yes | No* |

<sup>\*</sup>Non-compliant response; re-instruct in correct product usage procedure

<sup>\*\*</sup> Non-compliant response; exclude

# Signature Page for 300026 TMF- 238226 v 3.0

| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: PPD GMT+0000 |
|---|---|
| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: PPD GMT+0000 |
| Reason for signing: Approved | Name: PPD Role: Approver Date of signature: PPD GMT+0000 |

Signature Page for TMF-238226 v3.0